

# UNIVERSITY OF WASHINGTON SCHOOL OF MEDICINE FRED HUTCHINSON CANCER RESEARCH CENTER SEATTLE CANCER CARE ALLIANCE

**TITLE:** Phase II window study of pembrolizumab in untreated B-cell non-Hodgkin lymphoproliferative diseases

VERSION DATE: 21 July 2021

**VERSION NUMBER: 6.0** 

# **Investigator and Study Center:**

Sponsor-Investigator
Ajay K Gopal, MD
Professor, UW
Member, FHCRC
Seattle Cancer Care Alliance
825 Eastlake Ave. E. CE3-300
Seattle, WA 98109
Telephone: (206) 606-2037

This is an investigator-initiated study. The principal investigator Ajay Gopal, MD (who may also be referred to as the sponsor-investigator), is conducting the study and acting as the sponsor. Therefore, the legal/ethical obligations of the principal investigator include both those of a sponsor and those of an investigator.

FHCRC IRB Approval 03 16 2022 Document Released Date



# **TABLE OF CONTENTS**

| 1.0 | T | CRIAL SUMMARY 1 | 0 |
|-----|------|----------------------------------------------------------|---|
| 2.0 | T | TRIAL DESIGN | 0 |
| 2. | .1 | Trial Design | 0 |
| 2. | .2 | Trial Diagram1 | 0 |
| 3.0 | C | DBJECTIVE(S) & HYPOTHESIS(ES)1 | 1 |
| 3. | .1 | Primary Objective & Hypothesis 1 | 1 |
| 3. | .2 | Secondary Objectives & Hypotheses | 1 |
| 3. | .3 | Exploratory Objectives 1 | 1 |
| 4.0 | В | BACKGROUND & RATIONALE 1 | 1 |
| 4 | .1 | Background 1 | 1 |
| | 4.1. | Pembrolizumab: Pharmaceutical and Therapeutic Background | 2 |
| | 4.1. | 2 Preclinical and Clinical Trial Data | 3 |
| 4 | .2 | Rationale1 | 3 |
| | 4.2. | 1 Rationale for pembrolizumab in lymphoma | 3 |
| | 4.2. | 2 Rationale for Dose Selection/Regimen/Modification | 3 |
| | 4.2. | 3 Rationale for Endpoints | 5 |
| 5.0 | N | METHODOLOGY 1 | 5 |
| 5. | .1 | Entry Criteria1 | 5 |
| | 5.1. | 1 Diagnosis/Condition for Entry into the Trial | 5 |
| | 5.1. | 2 Subject Inclusion Criteria | 5 |
| | 5.1. | 3 Subject Exclusion Criteria | 7 |
| 5. | .2 | Trial Treatments1 | 8 |
| | 5.2. | 1 Dose Selection/Modification | 8 |



| 5.2.2 | Timing of Dose Administration | 20 |
|---|---|---|
| 5.3 | Concomitant Medications/Vaccinations (allowed & prohibited) | 20 |
| 5.3.1 | Acceptable Concomitant Medications | 20 |
| 5.3.2 | Prohibited Concomitant Medications. | 21 |
| 5.4 | Rescue Medications & Supportive Care | 21 |
| 5.4.1 | Supportive Care Guidelines | 21 |
| 5.5 | Diet/Activity/Other Considerations | 25 |
| 5.5.1 | Diet | 25 |
| 5.5.2 | Contraception | 25 |
| 5.5.3 | Use in Pregnancy | 25 |
| 5.5.4 | Use in Nursing Women | 26 |
| 5.6 | Subject Withdrawal/Discontinuation Criteria | 26 |
| <b>5.7</b> | Subject Replacement Strategy | 27 |
| 5.8 | Clinical Criteria for Early Trial Termination | 27 |
| 6.0 TF | RIAL FLOW CHART | 28 |
| 6.1 | Study Flow Chart | 28 |
| Adve | rse event assessment <sup>1</sup> | 28 |
| 7.0 TF | RIAL PROCEDURES | 29 |
| 7.1 | Trial Procedures | 29 |
| 7.1.1 | Administrative Procedures | 29 |
| 7.1.2 | Clinical Procedures/Assessments | 30 |
| 7.1.3 | Laboratory Procedures/Assessments | 33 |
| 7.1.4 | Other Procedures | 35 |
| 7.1.5 | Visit Requirements | 35 |
| 7.2 | Assessing and Recording Adverse Events | 36 |



| | , .2 | Definition of an Overdose for This Protocol and Reporting of Overdose to Merck | . 36 |
|---|---|---|---|
| | 7.2.2 | Reporting of Pregnancy and Lactation to the Sponsor and to Merck | . 37 |
| | 7.2.3 | Reporting of Adverse Events/Adverse Reactions | . 37 |
| | 7.2.4 | Evaluating Adverse Events | . 39 |
| | 7.2.5 | Sponsor-Investigator Responsibility for Reporting Adverse Events | . 42 |
| 8.0 | S | ΓATISTICAL ANALYSIS PLAN | . 43 |
| 8. | 1 | Statistical Analysis Plan Summary | . 43 |
| 8. | 2 | Statistical Analysis Plan | . 43 |
| 8. | 3 | Efficacy Analysis | . 44 |
| | 8.3.1 | Primary Efficacy Endpoint | . 44 |
| | 8.3.2 | 2 Secondary Efficacy Endpoints | . 44 |
| 9.0 | | ABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL UPPLIES | . 45 |
| 9. | 1 | Investigational Product | . 45 |
| 9.<br>9. | | Packaging and Labeling Information | |
| | 2 | | . 45 |
| 9. | 2 | Packaging and Labeling Information | . 45<br>. 46 |
| 9.<br>9. | 2<br>3<br>4 | Packaging and Labeling Information | . 45<br>. 46<br>. 46 |
| 9.<br>9.<br>9. | 2<br>3<br>4<br>5 | Packaging and Labeling Information | . 45<br>. 46<br>. 46 |
| 9.<br>9.<br>9.<br>10.0 | 2<br>3<br>4<br>5 | Packaging and Labeling Information Clinical Supplies Disclosure Storage and Handling Requirements Returns and Reconciliation | . 45<br>. 46<br>. 46<br>. 46 |
| 9.<br>9.<br>9.<br>10.0 | 2<br>3<br>4<br>5 | Packaging and Labeling Information Clinical Supplies Disclosure Storage and Handling Requirements Returns and Reconciliation DMINISTRATIVE AND REGULATORY DETAILS | . 45<br>. 46<br>. 46<br>. 46 |
| 9.<br>9.<br>9.<br>10.0<br>10 | 2<br>3<br>4<br>5<br>A | Packaging and Labeling Information Clinical Supplies Disclosure Storage and Handling Requirements Returns and Reconciliation DMINISTRATIVE AND REGULATORY DETAILS Data and Safety Monitoring Plan | . 45<br>. 46<br>. 46<br>. 46<br>. 46 |
| 9.<br>9.<br>9.<br>10.0<br>10 | 2<br>3<br>4<br>5<br>0.1<br>0.2<br>0.3 | Packaging and Labeling Information Clinical Supplies Disclosure Storage and Handling Requirements Returns and Reconciliation DMINISTRATIVE AND REGULATORY DETAILS Data and Safety Monitoring Plan Records | . 45<br>. 46<br>. 46<br>. 46<br>. 46<br>. 47 |
| 9.<br>9.<br>9.<br>10.0<br>10 | 2<br>3<br>4<br>5<br>A<br>0.1<br>0.2<br>0.3<br>EFE | Packaging and Labeling Information Clinical Supplies Disclosure Storage and Handling Requirements Returns and Reconciliation DMINISTRATIVE AND REGULATORY DETAILS Data and Safety Monitoring Plan Records Regulatory Responsibilities of Sponsor-Investigator | . 45<br>. 46<br>. 46<br>. 46<br>. 46<br>. 47<br>. 48 |



| 11.2 | Common Terminology Criteria for Adverse Events V4.0 (CTCAE) | 52 |
|---|---|---|
| 11.3 | Response Evaluation | 52 |
| 11 | 3.1 The Lugano Response Classification: For FL and MZL (21) | 52 |
| 11.4 | FLIPI Scoring System (26) | 55 |
| 11.5 | <b>Events of Clinical Interest Guidance Document: Version 5</b> | 56 |
| 11.9.1 0 | OVERVIEW | 56 |
| 3.1 | Pneumonitis | 58 |
| 3.2 | Colitis | 60 |
| 3.3 | Endocrine | 61 |
| 3.4 | Hematologic | 64 |
| 3.5 | Hepatic | 65 |
| 3.6 | Neurologic | 67 |
| <b>3.</b> 7 | Ocular | 67 |
| 3.8 | Renal | 68 |
| 3.9 | Skin | 69 |
| 3.10 | Immediate Evaluation for Potential Skin ECIs | 71 |
| 3.11 | Other | 72 |
| 3.12 | Infusion Reactions | 73 |
| 3.13 | Follow-up to Resolution | 74 |
| 5. Event | ts of Clinical Interest (ECI) – Reference Table | 74 |



## 1.0 TRIAL SUMMARY

| Abbreviated Title | Pembrolizumab in untreated indolent B-cell non-Hodgkin lymphoproliferative diseases |
|---|---|
| Trial Phase | II |
| Clinical Indication Indolent B-cell non-Hodgkin lymphoproliferative diseases without protection therapy | |
| Trial Type Nonrandomized, prospective trial | |
| Type of control | None |
| Route of administration | Intravenous |
| Treatment Groups Single group | |
| Number of trial subjects | 33 |
| Estimated enrollment period 18 months | |
| Estimated duration of trial | 36 months |
| Duration of participation 18 months | |

## 2.0 TRIAL DESIGN

# 2.1 Trial Design

This is a single arm phase II pilot study evaluating the efficacy of single-agent pembrolizumab for untreated, indolent B-cell non-Hodgkin lymphoproliferative diseases (iBCL) including follicular lymphoma (FL) and marginal zone lymphoma (MZL). In the window phase, treatment will be administered for up to six 3-week cycles and a response assessment performed at the conclusion. Patients that tolerate the drug and meet criteria for an objective response after 6 cycles may continue to receive pembrolizumab for up to an additional 12 cycles in the continuation phase. Patients who show progressive disease or stable disease after 6 cycles may be restaged after 3 additional cycles to assess for pseudoprogression/delayed response. Patients who show disease progression after 3 additional cycles will be removed from treatment. Patients who do not show evidence of disease progression may continue to receive pembrolizumab for up to a total of 18 cycles. A futility analysis will be performed after the first 5 subjects in each of two histologic subgroups (follicular lymphoma, marginal zone lymphoma) are treated. We anticipate that subjects will be enrolled over approximately 18 months and will be followed for outcomes for up to 5 years using standard-of-care assessments.



# 2.2 Trial Diagram



# 3.0 OBJECTIVE(S) & HYPOTHESIS(ES)

# 3.1 Primary Objective & Hypothesis

To gain a preliminary assessment of the efficacy of pembrolizumab as monotherapy for patients with untreated iBCL based on ORR measured at the end of a 6-cycle treatment period.

**Hypothesis:** Pembrolizumab will have an ORR of  $\geq$  50% in this untreated population after 6-cycles.

# 3.2 Secondary Objectives & Hypotheses

# (1) **Objective**:

To assess the safety and toxicity profile of pembrolizumab in patients with untreated iBCL.

**Hypothesis**: Pembrolizumab will not cause a significant degree of toxicity.

# (2) Objective:



To measure the efficacy of pembrolizumab used as monotherapy for patients with untreated iBCL by assessing clinical outcomes including complete response rate (CR), clinical benefit rate (CBR) defined as CR+partial response (PR)+ stable disease (SD)  $x \ge 6$  months, time to next therapy (TNT), progression-free survival (PFS), and the duration of response (DOR).

# 3.3 Exploratory Objectives

# (1) **Objectives:**

To evaluate clinical features including, as applicable, the follicular lymphoma international prognostic index (FLIPI) (see appendix 11.5), in addition to standard-of-care biomarkers including cytogenetics and Ki67 and correlate with response to pembrolizumab.

To evaluate baseline expression of proteins in the PD-1 pathway in archived tumor specimens and in pretreatment peripheral blood mononuclear cells and correlate with response to pembrolizumab.

To measure peripheral blood T-cell subsets and correlate with response to pembrolizumab.

## 4.0 BACKGROUND & RATIONALE

# 4.1 Background

B-cell non-Hodgkin lymphoproliferative diseases (BCL) are categorized according to how aggressively they behave. The indolent BCL subtypes (iBCL) include CLL/SLL, FL, MZL, WM/LPL, and, in some circumstances, MCL (1). Owing to immune activation, the early course of iBCL often is characterized by minimal progression or even spontaneous remission. The contribution of immune modulation in the natural history and treatment of iBCL has been borne out in preclinical studies (2) and early phase clinical trials (3-5).

iBCL inevitably relapse after therapy and typically become increasingly refractory to available treatments over time; iBCL are considered incurable short of allogeneic stem cell transplantation. Improving on this paradigm is necessary and requires novel strategies that minimize toxicity.

Anti-cancer therapies historically render the greatest benefit in the first-line treatment setting. This can be attributed to relatively undeveloped drug-resistance mechanisms in tumors and their smaller volume, in addition to the contribution of host immunity (6). The relatively slow early progression of iBCL makes this disease well suited to testing novel, low-toxicity treatment approaches in a predefined "window" of time (7).

# 4.1.1 Pembrolizumab: Pharmaceutical and Therapeutic Background

The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades (8). Accumulating evidence shows a correlation



between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies (9). In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated Tcells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2) (10). The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Pembrolizumab has recently been approved in the United Stated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilumumab and, if BRAF V600 mutation positive, a BRAF inhibitor.

## 4.1.2 Preclinical and Clinical Trial Data

Refer to the Investigator's Brochure for Preclinical and Clinical data.

## 4.2 Rationale

## 4.2.1 Rationale for pembrolizumab in lymphoma

As evidenced by the subset of patients with apparent spontaneous disease regression, the host immune system can play a significant role in iBCL (11, 12). Programmed cell death-1 (PD-1) is an immune checkpoint receptor expressed on activated T-cells. Tumor cells including lymphoid malignancies have been shown to express the ligands of PD-1: PD-L1 and PD-L2 (13). Engagement of T-cell PD-1 by its ligands downregulates T-cell activity through exhaustion. Modulation of the immune checkpoint pathway in iBCL has shown some promise in the relapsed and refractory setting in which the monoclonal PD-1 receptor blocking antibody nivolumab demonstrated activity as a single agent with an ORR in 4 of 10 patients treated in a phase I study (4). In a separate study the monoclonal anti-PD-1 antibody pidilizumab was combined with rituximab in patients with relapsed or refractory follicular lymphoma and



demonstrated an ORR in 19 or 29 patients (66%) with a median time to observed response of 88 days (range, 53 - 392) (5).

Pembrolizumab is a humanized monoclonal antibody of PD-1 with high affinity and potency. To date, pembrolizumab has shown an excellent safety and toxicity profile (see investigator's brochure), thereby fulfilling an important criterion for its use in the first-line window-of-opportunity setting (7). Use of immune checkpoint modulating antibodies as mono-therapy in the first-line setting has demonstrated efficacy in solid tumors (14, 15). Compared with the relapsed and refractory setting, untreated iBCL is accompanied by a relatively intact host immune repertoire with a potentially greater capacity to mount an effective anti-tumor immune response with immune-checkpoint inhibitor therapy.

## 4.2.2 Rationale for Dose Selection/Regimen/Modification

The choice of the 200 mg Q3W fixed dose is based on simulations performed using the population PK model of pembrolizumab showing that the fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.

A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage.

The first evaluation of the safety and pharmacokinetics of pembrolizumab was in an open-label Phase I trial (Protocol 001) conducted to evaluate the safety and clinical activity of single agent pembrolizumab. The dose escalation portion of this trial evaluated three dose levels, 1 mg/kg, 3 mg/kg, and 10 mg/kg, administered every 2 weeks (Q2W) in subjects with advanced solid tumors. All three dose levels were well tolerated and no dose-limiting toxicities were observed. This first in human study of pembrolizumab showed evidence of target engagement and objective evidence of tumor size reduction at all dose levels (1 mg/kg, 3 mg/kg and 10 mg/kg Q2W). No MTD has been identified to date. Recent data from other clinical studies within the pembrolizumab program has shown that a lower dose of pembrolizumab and a less frequent schedule may be sufficient for target engagement and clinical activity.

PK data analysis of pembrolizumab administered Q2W and Q3W showed slow systemic clearance, limited volume of distribution, and a long half-life (refer to IB). Pharmacodynamic data (IL-2 release assay) suggested that peripheral target engagement is durable (>21 days), providing scientific rationale for a Q3W dosing schedule.

A population pharmacokinetic analysis has been performed using serum concentration time data from 476 patients. Within the resulting population PK model, clearance and volume parameters of pembrolizumab were found to be dependent on body weight. The relationship between clearance and body weight, with an allometric exponent of 0.59, is within the range



observed for other antibodies and would support both body weight normalized dosing or a fixed dose across all body weights. Pembrolizumab has been found to have a wide therapeutic range based on the melanoma indication. The differences in exposure for a 200 mg fixed dose regimen relative to a 2 mg/kg Q3W body weight based regimen are anticipated to remain well within the established exposure margins of 0.5-5.0 for pembrolizumab in the melanoma indication. The exposure margins are based on the notion of similar efficacy and safety in melanoma at 10 mg/kg Q3W vs. the proposed dose regimen of 2 mg/kg Q3W (i.e. 5-fold higher dose and exposure). The population PK evaluation revealed that there was no significant impact of tumor burden on exposure. In addition, exposure was similar between the NSCLC and melanoma indications. Therefore, there are no anticipated changes in exposure between different indication settings.

The rationale for further exploration of 2 mg/kg and comparable doses including the fixed dose of 200 mg Q3W is based on: 1) similar efficacy and safety of pembrolizumab when dosed at either 2 mg/kg or 10 mg/kg Q3W in melanoma patients, 2) the flat exposure-response relationships of pembrolizumab for both efficacy and safety in the dose ranges of 2 mg/kg Q3W to 10 mg/kg Q3W, 3) the lack of effect of tumor burden or indication on distribution behavior of pembrolizumab (as assessed by the population PK model) and 4) the assumption that the dynamics of pembrolizumab target engagement will not vary meaningfully with tumor type.

# 4.2.3 Rationale for Endpoints

## 4.2.3.1 Efficacy Endpoints

Assessing the efficacy of pembrolizumab monotherapy in untreated iBCL will be performed according to standard response criteria (see section 7.2.1.5).

Because of the possibility of pseudoprogression(16), asymptomatic patients whose tumors demonstrate radiologic progression after initial restaging may receive therapy for 3 additional cycles and then will be restaged. Because of possibility of delayed response, patients whose tumors demonstrate stable disease may also receive therapy for 3 additional cycles and then will be restaged. Patients with tumor burden which doubles in size after initial restaging will be considered hyperprogression(17) and will not be eligible for the continuation stage.

## 4.2.3.2 Biomarker Research

Baseline expression by tumor cells and tumor-infiltrating cells of proteins involved in the PD-1 pathway will be performed on archived samples centrally when tissue is available; expression levels will be correlated with response to therapy.

Enumeration of peripheral blood T-cell subsets will be performed with flow cytometric evaluation of peripheral blood mononuclear cells before, during, and after treatment with pembrolizumab. These analyses will identify alterations in T-cell subsets as a possible biomarker predicting response to therapy.



## 5.0 METHODOLOGY

# 5.1 Entry Criteria

# 5.1.1 Diagnosis/Condition for Entry into the Trial

Patients must have a confirmed diagnosis of iBCL and not have received prior treatment for it. (Prior local radiotherapy is allowed as long as measurable disease is outside prior radiation field and all radiation-related adverse events have resolved.). Prior therapy that does not include any standard agents used for treatment of FL or MZL is also allowed as long as not in the same class of drugs as pembrolizumab.) Criteria for diagnosis include histopathologic evidence for FL and MZL.

# 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. Be willing and able to provide written informed consent/assent for the trial.
- 2. Be  $\geq$  18 years of age on day of signing informed consent.
- 3. Must have measurable disease defined by at least one of the following criteria:
  - a. Lesions greater than 1.5 cm that can be accurately measured in two dimensions by CT (preferred), or MRI.
- 4. Must have indication for treatment (Adapted from NCCN 2015 Guidelines)

Any of the following constitute an indication for treatment:

- a. Significant symptoms due to any iBCL: Which may include pain/discomfort, limitation of function, fatigue/malaise/constitutional symptoms, B-symptoms (fever, weight loss, night sweats), pruritus;
- b. Threatened end-organ function due to any iBCL;
- c. Progressive cytopenia secondary to any iBCL;
- d. Steady progression of FL and MZL
- 5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
- 6. Demonstrate adequate organ function as defined in Table 1.

Table 1 Adequate Organ Function Laboratory Values

| System | Laboratory Value |
|---------------------------------|----------------------------|
| Hematological | |
| Absolute neutrophil count (ANC) | ≥500/µL <sup>a, b</sup> |
| Platelets | ≥25 000/µL <sup>a, b</sup> |
| Hemoglobin | ≥8 g/dL <sup>a, b</sup> |
| Renal | |



| Creatinine OR Measured or calculated <sup>c</sup> creatinine clearance (GFR can also be used in place of creatinine or CrCl) | ≤1.5 × ULN <u>OR</u><br>≥30 mL/min for participant with creatinine levels<br>>1.5 × institutional ULN |
|---|---|
| Hepatic | |
| Total bilirubin | ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN |
| AST (SGOT) and ALT (SGPT) | ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) |
| Coagulation | |
| International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) | ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants |

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

- 7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
- 8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
- 9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

## 5.1.3 Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

- 1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
- 2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

<sup>&</sup>lt;sup>a</sup>Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed.

<sup>&</sup>lt;sup>b</sup>No lower limit if cytopenia is related to bone marrow involvement.

<sup>&</sup>lt;sup>c</sup>Creatinine clearance (CrCl) should be calculated per institutional standard.



- 3. Has a known history of active TB (Bacillus Tuberculosis).
- 4. Hypersensitivity to pembrolizumab or any of its excipients.
- 5. Has had prior chemotherapy, radiation therapy, or immunotherapy for the diagnosis of iBCL.
- 6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
- 7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
- 8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
- 9. Has known history of, or any evidence of active, non-infectious pneumonitis.
- 10. Has an active infection requiring systemic therapy.
- 11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
- 14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
- 15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
- 16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
- 17. Be in urgent need of therapy for lymphoma related complications (such as hyperviscosity syndrome) and those with bulky disease.
- 18. Has received a live vaccine within 30 days of planned start of study therapy.



Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

## **5.2** Trial Treatments

The treatment to be used in this trial is outlined below in **Table 2** 

**Table 2 Trial Treatment** 

| Drug | Dose/Potency | Dose<br>Frequency | Route of Administration | Regimen/Treatment<br>Period | Use |
|---|---|---|---|---|---|
| Pembrolizumab | 200 mg | Q3W | IV infusion | Day 1 of each 3<br>week cycle | Experimental |

## 5.2.1 Dose Selection/Modification

## **5.2.1.1** Dose Selection

The rationale for selection of the dose to be used in this trial is provided in Section 4.0 - Background and Rationale.

Details on preparation and administration of pembrolizumab are provided in the Pharmacy Manual.

## **5.2.1.2** Dose Modification

Adverse events (both non-serious and serious) associated with pembrolizumab exposure may represent an immunologic etiology. These adverse events may occur shortly after the first dose or several months after the last dose of treatment. Pembrolizumab must be withheld for drug-related toxicities and severe or life-threatening AEs as per Table 3 below. See Section 5.6.1 and Events of Clinical Interest Guidance Document for supportive care guidelines, including use of corticosteroids.



# Table 3 Dose Modification Guidelines for Drug-Related Adverse Events

# **General instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.
- **3.** For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with<br>corticosteroid and/or other<br>therapies | Monitor and follow-up |
|---|---|---|---|---|
| Pneumonitis | Grade 2 | Withhold | Administer corticosteroids (initial dose of 1-2 mg/kg prednisone or equivalent) followed by taper Add prophylactic antibiotics for | <ul> <li>Monitor participants for signs and symptoms of pneumonitis</li> <li>Evaluate participants with suspected pneumonitis with radiographic imaging and</li> </ul> |
| | Grade 3 or 4, or recurrent Grade 2 | Permanently discontinue | opportunistic infections | initiate corticosteroid treatment |
| Diarrhea / Colitis | Grade 2 or 3 | Withhold | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | Monitor participants for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus). |



| | Grade 4 or recurrent Grade 3 | Permanently discontinue | | <ul> <li>Participants with ≥ Grade 2 diarrhea suspecting colitis should consider GI consultation and performing endoscopy to rule out colitis.</li> <li>Participants with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion.</li> </ul> |
|---|---|---|---|---|
| AST / ALT<br>elevation or<br>Increased<br>bilirubin | Grade 2 <sup>a</sup> Grade 3 <sup>b</sup> or 4 <sup>c</sup> | Withhold Permanently discontinue | <ul> <li>Administer corticosteroids (initial dose of 0.5-1 mg/kg prednisone or equivalent) followed by taper</li> <li>Administer corticosteroids (initial dose of 1-2 mg/kg prednisone or equivalent) followed by taper</li> </ul> | Monitor with liver function tests (consider<br>weekly or more frequently until liver<br>enzyme value returned to baseline or is<br>stable |
| Type 1 diabetes<br>mellitus (T1DM)<br>or<br>Hyperglycemia | Newly onset<br>T1DM or<br>Grade 3 or 4<br>hyperglycemia<br>associated with<br>evidence of β-cell<br>failure | Withhold <sup>d</sup> | <ul> <li>Initiate insulin replacement<br/>therapy for participants with<br/>T1DM</li> <li>Administer anti-hyperglycemic in<br/>participants with hyperglycemia</li> </ul> | Monitor participants for hyperglycemia or other signs and symptoms of diabetes. |
| Hypophysitis | Grade 2 Grade 3 or 4 | Withhold or permanently discontinue <sup>d</sup> | Administer corticosteroids and initiate hormonal replacements as clinically indicated. | Monitor for signs and symptoms of<br>hypophysitis (including hypopituitarism and<br>adrenal insufficiency) |
| Hyperthyroidism | Grade 2 Grade 3 or 4 | Continue Withhold or permanently discontinue <sup>d</sup> | Treat with nonselective beta-<br>blockers (eg, propranolol) or<br>thionamides as appropriate | Monitor for signs and symptoms of thyroid disorders. |
| Hypothyroidism | Grade 2-4 | Continue | Initiate thyroid replacement<br>hormones (eg, levothyroxine or<br>liothyroinine) per standard of care | Monitor for signs and symptoms of thyroid disorders. |



| Nephritis grading<br>according to<br>increased<br>creatinine or<br>acute kidney<br>injury | Grade 2 Grade 3 or 4 | Withhold Permanently discontinue | Administer corticosteroids<br>(prednisone 1 to 2 mg/kg or<br>equivalent) followed by taper. | • | Monitor changes of renal function |
|---|---|---|---|---|---|
| Neurological<br>Toxicities | Grade 3 or 4 | Permanently discontinue | Based on severity of AE administer corticosteroids | • | Ensure adequate evaluation to confirm etiology and/or exclude other causes |
| Myocarditis | Grade 1 | Withhold | Based on severity of AE administer corticosteroids | • | Ensure adequate evaluation to confirm etiology and/or exclude other causes |
| | Grade 2, 3 or 4 | Permanently discontinue | | | |
| Exfoliative<br>Dermatologic | Suspected SJS,<br>TEN, or DRESS | Withhold | Based on severity of AE administer corticosteroids | • | Ensure adequate evaluation to confirm etiology or exclude other causes |
| Conditions | Confirmed SJS,<br>TEN, or DRESS | Permanently discontinue | | | |
| All other irAEs | Persistent Grade 2 | Withhold | Based on type and severity of AE administer corticosteroids | • | Ensure adequate evaluation to confirm etiology and/or exclude other causes |
| | Grade 3 | Withhold or discontinue based on the type of event <sup>e</sup> . | | | |
| | Grade 4 or recurrent Grade 3 | Permanently discontinue | | | |

AE(s)=adverse event(s); ALT= alanine aminotransferase; AST=aspartate aminotransferase; CTCAE=Common Terminology Criteria for Adverse Events; DRESS=Drug Rash with Eosinophilia and Systemic Symptom; GI=gastrointestinal; IO=immuno-oncology; ir=immune related; IV=intravenous; SJS=Stevens-Johnson Syndrome; T1DM=type 1 diabetes mellitus; TEN=Toxic Epidermal Necrolysis; ULN=upper limit of normal.

# Note: Non-irAE will be managed as appropriate, following clinical practice recommendations.

- <sup>a</sup> AST/ALT: >3.0 to 5.0 x ULN if baseline normal; >3.0 to 5.0 x baseline, if baseline abnormal; bilirubin:>1.5 to 3.0 x ULN if baseline normal; >1.5 to 3.0 x baseline if baseline abnormal
- b AST/ALT: >5.0 to 20.0 x ULN, if baseline normal; >5.0 to 20.0 x baseline, if baseline abnormal; bilirubin:>3.0 to 10.0 x ULN if baseline normal; >3.0 to 10.0 x baseline abnormal
- <sup>c</sup> AST/ALT: >20.0 x ULN, if baseline normal; >20.0 x baseline, if baseline abnormal; bilirubin: >10.0 x ULN if baseline normal; >10.0 x baseline if baseline abnormal
- d The decision to withhold or permanently discontinue pembrolizumab is at the discretion of the investigator or treating physician. If control achieved or ≤ Grade 2, pembrolizumab may be resumed.



| e | Events that require discontinuation include, but are not limited to: encephalitis and other clinically important irAEs (e.g., vasculitis and sclerosing cholangitis). |
|---|---|

Dosing interruptions are permitted in the case of medical / surgical events or logistical reasons not related to study therapy (e.g., elective surgery, unrelated medical events, patient vacation, and/or holidays). Subjects should be placed back on study therapy within 3 weeks of the scheduled interruption, unless otherwise discussed with the Sponsor-Investigator or lead sub-investigator. The reason for interruption should be documented in the patient's study record.



# **5.2.2** Timing of Dose Administration

Trial treatment should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6.0). Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial treatments will be administered on an outpatient basis.

Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

The Pharmacy Manual contains specific instructions for the preparation of the pembrolizumab infusion fluid and administration of infusion solution.

# 5.3 Concomitant Medications/Vaccinations (allowed & prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The sponsor-investigator should discuss any questions regarding this with the Merck Clinical team. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician.

## 5.3.1 Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the case report form (CRF) including all prescription, over-the-counter (OTC), herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the CRF.

All concomitant medications received within 28 days before the first dose of trial treatment and 30 days after the last dose of trial treatment should be recorded. Concomitant medications administered after 30 days after the last dose of trial treatment should be recorded for SAEs and ECIs as defined in Section 7.2.

## **5.3.2** Prohibited Concomitant Medications

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post response/stable disease relapse) of this trial:



- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol
- Chemotherapy not specified in this protocol
- Investigational agents other than pembrolizumab
- Radiation therapy
- Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.
- Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor-investigator.

Subjects who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describes other medications which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

## **5.4** Rescue Medications & Supportive Care

# **5.4.1** Supportive Care Guidelines

Subjects should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of adverse events with potential immunologic etiology are outlined below and in greater detail in the ECI guidance document. Where appropriate, these guidelines include the use of oral or intravenous treatment with corticosteroids as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the investigator determines the events to be related to pembrolizumab.

Note: if after the evaluation the event is determined not to be related, the investigator is instructed to follow the ECI reporting guidance but does not need to follow the treatment guidance (as outlined in the ECI guidance document). Refer to Section 5.2.1 for dose modification.

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event. Suggested conditional procedures, as appropriate, can be found in the ECI guidance document.



#### • Pneumonitis:

- For Grade 2 events, treat with systemic corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- o For **Grade 3-4 events**, immediately treat with intravenous steroids. Administer additional anti-inflammatory measures, as needed.
- Add prophylactic antibiotics for opportunistic infections in the case of prolonged steroid administration.

#### • Diarrhea/Colitis:

Subjects should be carefully monitored for signs and symptoms of enterocolitis (such as diarrhea, abdominal pain, blood or mucus in stool, with or without fever) and of bowel perforation (such as peritoneal signs and ileus).

- O All subjects who experience diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion. For Grade 2 or higher diarrhea, consider GI consultation and endoscopy to confirm or rule out colitis.
- o For **Grade 2 diarrhea/colitis** that persists greater than 3 days, administer oral corticosteroids.
- o For **Grade 3 or 4 diarrhea/colitis** that persists > 1 week, treat with intravenous steroids followed by high dose oral steroids.
- o When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

# • Type 1 diabetes mellitus (if new onset, including diabetic ketoacidosis [DKA]) or ≥ Grade 3 Hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA)

## o For **T1DM** or **Grade 3-4** Hyperglycemia

- Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
- Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.

# • Hypophysitis:

- For Grade 2 events, treat with corticosteroids. When symptoms improve to Grade
  1 or less, steroid taper should be started and continued over no less than 4 weeks.
  Replacement of appropriate hormones may be required as the steroid dose is
  tapered.
- o For **Grade 3-4** events, treat with an initial dose of IV corticosteroids followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper



should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

# • Hyperthyroidism or Hypothyroidism:

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.

- o Grade 2 hyperthyroidism events (and Grade 2-4 hypothyroidism):
  - In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
  - In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- o **Grade 3-4** hyperthyroidism
  - Treat with an initial dose of IV corticosteroid followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

## • Hepatic:

- o For **Grade 2** events, monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with IV or oral corticosteroids
- o For **Grade 3-4** events, treat with intravenous corticosteroids for 24 to 48 hours.
- o When symptoms improve to Grade 1 or less, a steroid taper should be started and continued over no less than 4 weeks.

# • Renal Failure or Nephritis:

- o For **Grade 2** events, treat with corticosteroids.
- o For Grade 3-4 events, treat with systemic corticosteroids.
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- **Management of Infusion Reactions**: Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Table 4 below shows treatment guidelines for subjects who experience an infusion reaction associated with administration of pembrolizumab.

**Table 4 Infusion Reaction Treatment Guidelines** 



| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |
| Grade 2 Requires infusion interruption but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for < =24 hrs | Stop Infusion and monitor symptoms. Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDs Acetaminophen Narcotics Increase monitoring of vital signs as medically indicated until the participant is deemed medically stable in the opinion of the investigator. If symptoms resolve within 1 hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate (e.g. from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the participant should be premedicated for the next scheduled dose. Subjects who develop Grade 2 toxicity despite adequate premedication should be permanently discontinued from further trial | Subject may be premedicated 1.5f (± 30 minutes) prior to infusion of pembrolizumab (PEMBROLIZUMAB) with: Diphenhydramine 50 mg po (or equivalent dose of antihistamine). Acetaminophen 500-1000 mg po (or equivalent dose of antipyretic) |
| Grades 3 or 4 | treatment administration. Stop Infusion. | No subsequent dosing |
| Grade 3: Prolonged (i.e., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for other clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDS Acetaminophen Narcotics Oxygen Pressors Corticosteroids Epinephrine** | Tro subsequent dosing |
| Grade 4:<br>Life-threatening; pressor or ventilatory<br>support indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. Hospitalization may be indicated. **In cases of anaphylaxis, epinephrine should be used immediately. Subject is permanently discontinued from further trial treatment administration. ould be available in the room and a physician readily | |

# 5.5 Diet/Activity/Other Considerations

# 5.5.1 Diet

Subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.



## 5.5.2 Contraception

Pembrolizumab may have adverse effects on a fetus in utero. Furthermore, it is not known if pembrolizumab has transient adverse effects on the composition of sperm. Non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive. Highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is ≥45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from study Visit 1 throughout the study period up to 120 days after the last dose of study therapy.

The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

Subjects should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study. In order to participate in the study, they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period defined in section 7.2.2-Reporting of Pregnancy and Lactation to the Sponsor-Investigator and to Merck. If there is any question that a subject will not reliably comply with the requirements for contraception, that subject should not be entered into the study.

## 5.5.3 Use in Pregnancy

If a subject inadvertently becomes pregnant while on treatment with pembrolizumab, the subject will immediately be removed from the study. The site will contact the subject at least monthly and document the subject's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to to Merck without delay and within 24 hours to the Sponsor-Investigator and within 2 business days of investigator knowledge if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn).

The study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to Merck. If a male subject impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported to Merck and followed as described above and in Section 7.2.2.

## 5.5.4 Use in Nursing Women

It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, subjects who are breast-feeding are not eligible for enrollment.



# 5.6 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons. Subjects who require cessation of study therapy but do not withdraw consent may remain in standard follow-up for up to 5 years.

A subject must be discontinued from the trial for any of the following reasons:

- The subject or legal representative (such as a parent or legal guardian) withdraws consent.
- Confirmed radiographic disease progression
- Unacceptable adverse experiences as described in Section 5
- Intercurrent illness that prevents further administration of treatment
- Investigator's decision to withdraw the subject
- The subject has a confirmed positive serum pregnancy test
- Noncompliance with trial treatment or procedure requirements
- The subject is lost to follow-up
- Administrative reasons

The End of Treatment and Follow-up visit procedures are listed in Section 6 (Protocol Flow Chart) and Section 7.1.5 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events may be collected for 90 days after the end of treatment as described in Section 7.2.3.1). Patients may have post-treatment follow-up for disease status up to 5 years at longest, or until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up.

## 5.7 Subject Replacement Strategy

Subjects who fail to complete study therapy will not be replaced.

# 5.8 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

- 1. Quality or quantity of data recording is inaccurate or incomplete
- 2. Poor adherence to protocol and regulatory requirements



- 3. Incidence or severity of adverse drug reaction in this or other studies indicates a potential health hazard to subjects
- 4. Plans to modify or discontinue the development of the study drug

In the event of Merck decision to no longer supply study drug, ample notification will be provided so that appropriate adjustments to subject treatment can be made.

## 6.0 TRIAL FLOW CHART

## 6.1 Study Flow Chart

| | Screening<br>Period | Treatment Phase | | End of treatment <sup>6</sup> | Long-term<br>Follow-up <sup>7</sup> | |
|---|---|---|---|---|---|---|
| | | Window<br>Cycles (1-6) | Response assessment <sup>8</sup> | Continuation Cycles (7-18)9 | | • |
| Scheduling and Timing | -42 to -1d | +/- 3d | | +/- 3d | | |
| Informed consent | X | | | | | |
| Inclusion/Exclusion criteria | X | | | | | |
| Medical history | X | | | | | |
| Medication review (prior and concomitant) | X | X | | X | | |
| Trial treatment administration | | X | | X | | |
| Post-study anticancer therapy status | | | | | | X |
| Survival status | | | | | | X |
| Vital signs | X | X | | X | X | |
| Physical exam | X | X | | X | X | |
| ECOG performance status | X | X | | X | X | |
| Adverse event assessment <sup>1</sup> | X | X | | X | X | |
| CBC and differential | X | X | X | X | X | |
| Comprehensive metabolic panel and LDH | X | X | X | X | X | |
| HepB SAg, Hep B Core Ab,<br>HepC Antibody and HIV screen | X | | | | | |
| Urinalysis | X | | | | | |
| T3, FT4, and TSH | X | X | | X | X | |
| PT/INR and aPTT | X | | | | | |
| Correlative studies blood draw | X | | X | | X | |
| Bone marrow studies <sup>2</sup> | X | | | | X | |
| Pregnancy test <sup>3</sup> | X | | | | | |
| Tumor assessment <sup>5</sup> | X | X | X | X | X | |
| Archival Tissue collection <sup>4</sup> | X | | | | | |

<sup>&</sup>lt;sup>1</sup>Adverse events will be recorded from the time of a subject signing consent up until 30 days after the last dose of pembrolizumab, or 90 days after the last dose of pembrolizumab in the case of serious adverse events.

<sup>&</sup>lt;sup>2</sup>If bone marrow involvement by iBCL was previously shown then repeat bone marrow exam at screening is not required as it is assumed positive. Otherwise, bone marrow studies include aspirate and unilateral biopsy and should be performed at screening unless a waiver is approved by the study Sponsor-Investigator or sub-Investigator. If all bone marrow studies are negative at screening, these do not need to be repeated. If bone marrow status is unknown or positive at screening, patients will need to a have bone marrow study for confirmation of a CR.

<sup>&</sup>lt;sup>3</sup> Pregnancy test is only required in women of childbearing potential.

<sup>&</sup>lt;sup>4</sup>Archived tumor samples are requested for pathologic confirmation and biomarker analysis. If an archived specimen is not available or contains insufficient material, a fresh tumor biopsy (if clinically feasible) will be requested. Correlative studies may be performed on any available tissue.

<sup>&</sup>lt;sup>5</sup>Tumor assessment labs and/or imaging (see section 7.1.2.5) will be performed prior to cycle 4 (within 7 days of scheduled treatment dose) during the window phase. Tumor assessment will be performed prior to cycle 7 (within 7 days of scheduled treatment dose) to determine eligibility for continuation on study in continuation phase. Tumor assessment labs and/or imaging will be performed prior to cycles 11 and 15 (within 7 days of scheduled treatment dose) during the continuation phase, as applicable. Tumor assessment labs and/or imaging will be performed at end-of-treatment evaluation only for subjects who did not have tumor assessment labs and/or imaging performed within 60 days of end-of-treatment. Tumor assessment labs and/or imaging will also be performed as indicated per clinical standard of care (e.g. as appropriate for disease, to evaluate clinical suspicion of disease progression). Patients who have stable disease or asymptomatic radiologic disease progression prior to cycle 7 will remain in the window phase with restaging prior to cycle 10 to evaluate for pseudoprogression or delayed response. Patients who have restaging prior to cycle 10 are not required to have tumor assessments prior to cycle 11. Patients who have radiologic disease progression with doubling of tumor size prior to cycle 7 will be categorized as hyperprogression and will not proceed to the continuation phase.

<sup>&</sup>lt;sup>6</sup>End-of-treatment evaluations should be done within 30 days (+/- 14 days) of the last dose of pembrolizumab or prior to the start of a new anti-cancer drug, whichever is first.

<sup>&</sup>lt;sup>7</sup>Long-term follow-up should be done according to the patient's physician standard of care. This may be performed at patients' local physician's offices. Long-term follow-up will assess survival and disease progression; for clarification, subjects may be contacted by the study team until death, subject withdrawal of consent, lost to follow-up, or study termination, whichever occurs first.

<sup>&</sup>lt;sup>8</sup>Response assessment will be performed prior to cycle 7 (within 7 days of scheduled treatment dose) only for those subjects that complete 6 cycles of treatment in the window phase.

<sup>9</sup>During treatment in the continuation phase, clinical assessment (physical exam including performance status, adverse event and medication review) will be performed on day 1 (+/- 3 days) of each odd-numbered cycle only, or as clinically indicated. Studies performed for response assessment on to end to be repeated prior to cycle 7.

#### 7.0 TRIAL PROCEDURES

## 7.1 Trial Procedures

The Trial Flow Chart in Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the investigator and/or Merck for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

## 7.1.1 Administrative Procedures

## 7.1.1.1 Informed Consent

The investigator must obtain documented consent from each potential subject prior to participating in a clinical trial.

#### 7.1.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements and applicable laws and regulations.

## 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial.

# 7.1.1.3 Medical History

A medical history will be obtained by the investigator or qualified designee. Medical history will include all active conditions, and any condition diagnosed within the prior 10 years that are considered to be clinically significant by the investigator. Details regarding the disease for which the subject has enrolled in this study will be recorded separately and not listed as medical history.

## 7.1.1.4 Prior and Concomitant Medications Review

## 7.1.1.4.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the subject within 28 days before starting the trial. The subject will not have received prior treatment for the disease.

#### 7.1.1.4.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial. All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

## 7.1.1.5 Disease Details and Treatments

## 7.1.1.5.1 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

# 7.1.1.5.2 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-neoplastic therapy initiated after the last dose of trial treatment.

# 7.1.2 Clinical Procedures/Assessments

# 7.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart and more frequently if clinically indicated. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 4.0 (see Section 11.2). Toxicities will be

characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

For subjects receiving treatment with pembrolizumab all AEs of unknown etiology associated with pembrolizumab exposure should be evaluated to determine if it is possibly an event of clinical interest (ECI) of a potentially immunologic etiology (termed immune-related adverse events, or irAEs); see the separate ECI guidance document in Appendix 11.3.10 regarding the identification, evaluation and management of potential irAEs.

Please refer to section 7.2 for detailed information regarding the assessment and recording of AEs.

# 7.1.2.2 Physical Exam

The investigator or qualified designee will perform a complete physical exam during the screening period. Clinically significant abnormal findings should be recorded as medical history. A physical exam should be performed during screening.

# **7.1.2.3 Vital Signs**

Vital signs will be taken at screening, prior to the administration of each dose of trial treatment and at treatment discontinuation as specified in the Trial Flow Chart (Section 6.0). Vital signs should include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.

# 7.1.2.4 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (see Section 11.1) at screening, prior to the administration of trial treatment, and after discontinuation of trial treatment as specified in the Trial Flow Chart.

## 7.1.2.5 Tumor Imaging and Assessment of Disease

Tumor imaging and assessment of disease will be performed according to each disease subtype:

## 7.1.2.5.1 Follicular lymphoma

FDG-PET imaging will be required during study screening and prior to treatment on cycle 7 to determine candidacy for continuation on study. Contrast-enhanced computed tomography (CT) of the chest, abdomen, and pelvis alone will be performed at each tumor assessment. For measurement of response, 2014 criteria as described in "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification" will be used (see Appendix 11.3.1) (18). CT imaging of the neck will be performed as indicated for standard of care.

All CT scans should be performed with IV contrast unless contraindicated, and abdominal and pelvis scans should be performed with oral contrast.

# 7.1.2.5.2 Marginal Zone Lymphoma in which Nodal Disease is Known or Suspected

CT of the chest, abdomen, and pelvis will be performed at each tumor assessment. For measurement of response, 2014 criteria as described in "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification" will be used (see Appendix 11.3.2) (18). CT imaging of the neck will be performed as indicated for standard of care.

All CT scans should be performed with IV contrast unless contraindicated, and abdominal and pelvis scans should be performed with oral contrast.

# 7.1.2.6 Bone marrow aspirate and biopsy

A bone marrow aspirate and biopsy will be obtained before the first dose of study drug, and for confirmation of CR when indicated. Bone marrow aspirate and biopsy requirements may be waived by the Sponsor-Investigator or lead sub-Investigator. These samples will be evaluated locally.

# 7.1.2.7 Tumor Tissue Collection and Correlative Studies Blood Sampling

Assessment of available archived tumor tissue for correlative study analysis will be performed during the screening period. Available pretreatment biopsy tissue will be provided for correlative study analysis. Peripheral blood correlative study samples will be collected during screening, at response assessment, and at end-of-treatment (see Section 6.1).

# Specimen Requirements

- A 5-10 mL specimen of peripheral blood in a lavender- (EDTA) or green- (sodium heparin) tube is acceptable for each draw.
- Storage/Transport Temperature: Specimens can be transported with a cold pack or wet ice, but do not fix or freeze specimens.
- Unacceptable Conditions: Frozen specimens, specimens greater than 48 hours old, specimens fixed in formalin for flow cytometry.

## Address for shipping specimens:

Seattle Cancer Care Alliance Hematopathology Laboratory G7800 825 Eastlake Ave E. Seattle, WA 98109

# 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below and in Section 6.1. All chemistry and hematology studies may be performed within 3 days of pembrolizumab dosing prior to day 1 of each cycle.

Laboratory tests for hematology, chemistry, urinalysis, and others are specified in Table 5.

Table 5 Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Serum β-human chorionic gonadotropin† |
| Hemoglobin | Alkaline phosphatase | Glucose | (β-hCG)† |
| Platelet count | Alanine aminotransferase (ALT) | Protein | PT (INR) |
| WBC (total and differential) | Aspartate aminotransferase (AST) | Specific gravity | aPTT |
| Red Blood Cell Count | Lactate dehydrogenase (LDH) | Microscopic exam (If abnormal) | Total thriiodothyronine (T3) |
| Absolute Neutrophil Count | Carbon Dioxide ‡ | results are noted | Free tyroxine (T4) |
| Absolute Lymphocyte Count | (CO <sub>2</sub> or biocarbonate) | Urine pregnancy test † | Thyroid stimulating hormone (TSH) |
| | Uric Acid | | Hepatitis B Surface Antigen (HBsAg) |
| | Calcium | | Hepatitis B Core Antibody (HBcAb) |
| | Chloride | | Hepatitis C Antibody |
| | Glucose | | HIV Screening |
| | Phosphorus | | PK |
| | Potassium | | Blood for correlative studies |
| | Sodium | | |
| | Magnesium | | |
| | Total Bilirubin | | |
| | Direct Bilirubin (If total bilirubin is elevated above the upper limit of normal) | | |
| | Total protein | | |
| | Blood Urea Nitrogen | | |

<sup>†</sup> Perform on women of childbearing potential only. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test will be required.


<sup>‡</sup> If considered standard of care in your region.

Results must be reviewed by the investigator or qualified designee and found to be acceptable prior to each dose of trial treatment.

## 7.1.4 Other Procedures

## 7.1.4.1 Withdrawal/Discontinuation

When a subject discontinues/withdraws prior to trial completion, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events.

# 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

## **7.1.5.1** Screening

## 7.1.5.1.1 Screening Period

The screening period begins upon signing consent and includes evaluations as described in Section 6.1. The screening period may last up to 42 days.

## 7.1.5.2 Treatment Period

The treatment period includes the window phase during which pembrolizumab is administered every 21 (+/- 3) days for 6 cycles. Subjects that are determined to have an objective response or stable disease at the point of response assessment prior to cycle 7 (or cycle 10 if pseudoprogression/delayed response) may continue on study in the continuation phase. During the continuation phase pembrolizumab is administered every 21 (+/- 3) days for up to 12 additional cycles to complete a total of up to 18 cycles.

## 7.1.5.3 End-of-treatment Visit

Thirty days (+/- 14 d) after the last dose of pembrolizumab, irrespective of cause of cessation, an end-of-treatment visit should be performed. However, if a subject requires additional anti-cancer therapy, the off-study visit may occur earlier.

The off-study visit will include laboratory studies, medical history, physical exam, remission status, concomitant medications, adverse events, and documentation of any ECI and subsequent management, as in Section 6.0. All AEs that occur prior to the end-of-treatment visit should be recorded. Subjects with an AE of Grade > 1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-neoplastic therapy, whichever occurs first. SAEs that occur within 90 days of the end of treatment or before initiation of a new anti-cancer treatment should also be followed and recorded.
After the end-of-study visit, additional follow-up will be conducted as per routine standard of care for up to 5 years unless other criteria for withdrawal are met (see Section 5.6). Long-term follow-up may be performed at patients' local physician's offices. Long-term follow-up will assess survival and disease progression; for clarification, subjects may be contacted by the study team until death, subject withdrawal of consent, lost to follow-up, or study termination, whichever occurs first.

## 7.2 Assessing and Recording Adverse Events

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Merck's product, is also an adverse event.

Merck product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by Merck for human use.

Adverse events may occur during the course of the use of Merck product in clinical trials or within the follow-up period specified by the protocol, or prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

Adverse events may also occur in screened subjects during any pre-allocation baseline period as a result of a protocol-specified intervention, including washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

Progression of the cancer under study is not considered an adverse event unless it is considered to be drug related by the investigator.

Adverse events grade 3 and higher, as well as AEs requiring clinical intervention/dose modification, ECIs and SAEs of any grade, will be recorded from the time the consent form is signed up until 90 days following the last dose of pembrolizumab and at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1.

## 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to Merck

For purposes of this trial, an overdose of pembrolizumab will be defined as any dose of 1,000 mg or greater ( $\geq$ 5 times the indicated dose). No specific information is available on the treatment of overdose of pembrolizumab. Appropriate supportive treatment should be provided if clinically indicated. In the event of overdose, the subject should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

If an adverse event(s) is associated with ("results from") the overdose of a Merck product, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Merck's product meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

All reports of overdose with and without an adverse event must be reported within 2 working days of investigator knowledge to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

## 7.2.2 Reporting of Pregnancy and Lactation to the Sponsor and to Merck

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them), including the pregnancy of a male subject's female partner that occurs during the trial or within 120 days of completing the trial completing the trial, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. All subjects and female partners of male subjects who become pregnant must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

Such events must be reported within 2 working days of investigator knowledge to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

## 7.2.3 Reporting of Adverse Events/Adverse Reactions

#### 7.2.3.1 Serious Adverse Events

A serious adverse event is any adverse event occurring at any dose or during any use of Merck's product that:

- Results in death;
- Is life threatening;
- Results in persistent or significant disability/incapacity;
- Results in or prolongs an existing inpatient hospitalization;
- Is a congenital anomaly/birth defect;
- Is a new cancer (that is not a condition of the study);
- Is associated with an overdose;
- Is an other important medical event

Refer to Table 6 for additional details regarding each of the above criteria.

Any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study that occurs to any subject from the time the consent is signed through 90 days following cessation of treatment, or the initiation of new anti-cancer therapy, whichever is earlier, whether or not related to Merck product, must be reported within 2 business days of investigator knowledge to Merck Global Safety.

Non-serious Events of Clinical Interest will be forwarded to Merck Global Safety and will be handled in the same manner as SAEs.

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to Merck product that is brought to the attention of the investigator at any time outside of the time period specified in the previous paragraph also must be reported immediately to Merck.

# SAE reports and any other relevant safety information are to be forwarded to the Merck Global Safety facsimile number: +1-215-993-1220

A copy of all 15 Day Reports and Annual Progress Reports is submitted as required by FDA, Pharmaceutical and Medical Devices agency (PMDA) or other local regulators. Investigators will cross reference this submission according to local regulations to the Merck Investigational Compound Number (IND, CSA, etc.) at the time of submission. Additionally, investigators will submit a copy of these reports to Merck & Co., Inc. (Attn: Worldwide Product Safety; FAX 215 993-1220) at the time of submission to FDA.

All subjects with serious adverse events must be followed up for outcome.

#### 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI). See appendix 11.10, ECI Guidance Document, for management and reporting of ECI. ECI and must be recorded as such on the Adverse Event case report forms/worksheets and reported within 2 business days of investigator knowledge to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220) Events of clinical interest for this trial include:

- 1. An overdose of Merck product, as defined in Section 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to Merck, that is not associated with clinical symptoms or abnormal laboratory results.
- 2. An elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing. \*

\*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology. The trial site guidance for assessment and follow up of these criteria can be found in the Investigator Trial File Binder (or equivalent).

## 1. Additional adverse events:

A separate guidance document has been provided entitled "Event of Clinical Interest Guidance Document" (previously entitled, "Event of Clinical Interest and Immune-Related Adverse Event Guidance Document"). This document can be found in Appendix 4 and provides guidance regarding identification, evaluation and management of ECIs and irAEs.

ECIs (both non-serious and serious adverse events) identified in this guidance document from the date of first dose through 90 days following cessation of treatment, or 30 days after the initiation of a new anticancer therapy, whichever is earlier, need to be reported within 2 business days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220), regardless of attribution to study treatment, consistent with standard SAE reporting guidelines.

Subjects should be assessed for possible ECIs prior to each dose. Lab results should be evaluated and subjects should be asked for signs and symptoms suggestive of an immune-related event. Subjects who develop an ECI thought to be immune-related should have additional testing to rule out other etiologic causes. If lab results or symptoms indicate a possible immune-related ECI, then additional testing should be performed to rule out other etiologic causes. If no other cause is found, then it is assumed to be immune-related.

## 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 4.0. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

All adverse events regardless of CTCAE grade must also be evaluated for seriousness.

## Table 6 Evaluating Adverse Events

An investigator who is a qualified physician, will evaluate all adverse events as to:

| V4.0 CTCAE<br>Grading | Grade 1 Mild; asymptomatic or mid symptoms; clinical or diagnostic observations only; intervention not indicated. | |
|---|---|---|
| J | Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. |
| | Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation or hospitalization indicated; |
| | | disabling; limiting self-care ADL. |
| | Grade 4 | Life threatening consequences; urgent intervention indicated. |
| | Grade 5 | Death related to AE |
| Seriousness | A serious adverse e | event is any adverse event occurring at any dose or during any use of Merck product that: |
| | †Results in death; | |
| | †Is life threatening | g; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an |
| | adverse event that, | had it occurred in a more severe form, might have caused death.); or |
| | †Results in a persi | stent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or |
| | †Results in or pro | longs an existing inpatient hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay, even if the |
| | | precautionary measure for continued observation. (Note: Hospitalization [including hospitalization for an elective procedure] for a preexisting |
| | | s not worsened does not constitute a serious adverse event.); or |
| | †Is a congenital ar | nomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis);or |
| | | hat is not a condition of the study) or |
| | Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event. An overdose that is not | |
| | associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, | |
| | | based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes |
| | listed previously (designated above by a †). | |
| Duration | | Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units |
| Action taken | Did the adverse event cause the Merck product to be discontinued? | |
| Relationship to | Did the Merck product cause the adverse event? The determination of the likelihood that the Merck product caused the adverse event will be provided by an | |
| test drug | investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE | |
| | | medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The |
| | criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event | |
| | based upon the ava | |
| | | aponents are to be used to assess the relationship between the Merck product and the AE; the greater the correlation with the components and |
| | their respective elements (in number and/or intensity), the more likely the Merck product caused the adverse event (AE): | |
| | Exposure | Is there evidence that the subject was actually exposed to the Merck product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? |
| | Time Course | Did the AE follow in a reasonable temporal sequence from administration of the Merck product? |
| | | Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? |
| | Likely Cause Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other factors | |


| Relationship | The following components are to be used to assess the relationship between the test drug and the AE: (continued) | |
|---|---|---|
| to Merck | Dechallenge | Was the Merck product discontinued or dose/exposure/frequency reduced? |
| product | | If yes, did the AE resolve or improve? |
| (continued) | | If yes, this is a positive dechallenge. If no, this is a negative dechallenge. |
| | (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE resolved/impro | |
| | | of the Merck product; or (3) the trial is a single-dose drug trial); or (4) Merck product(s) is/are only used one time.) |
| | Rechallenge | Was the subject re-exposed to the Merck product in this study? |
| | | If yes, did the AE recur or worsen? |
| | | If yes, this is a positive rechallenge. If no, this is a negative rechallenge. |
| | | (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) the trial is a single-dose drug trial); or |
| | | (3) Merck product(s) is/are used only one time). |
| | | NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS AND WHICH MAY HAVE BEEN |
| | | CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES ADDITIONAL POTENTIAL |
| | | SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN ADVANCE BY THE U.S. CLINICAL |
| | | MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. |
| | Consistency | Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Merck product or drug class pharmacology |
| with Trial or toxicology? | | or toxicology? |
| | Treatment | |
| | Profile | |
| | f relationship will be<br>he above elements. | e reported on the case report forms /worksheets by an investigator who is a qualified physician according to his/her best clinical judgment, including |
| Record one of th | e following | Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Merck product relationship). |
| Yes, there is a reasonable possibility of Merck product relationship. | | There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the administration of the Merck product is reasonable. The AE is more likely explained by the Merck product than by another cause. |
| No, there is not a possibility Mercl relationship | | Subject did not receive the Merck product OR temporal sequence of the AE onset relative to administration of the Merck product is not reasonable OR there is another obvious cause of the AE. (Also entered for a subject with overdose without an associated AE.) |


## 7.2.5 Sponsor-Investigator Responsibility for Reporting Adverse Events

The sponsor-investigator is required to report all problems, events and information that require prompt reporting to the IRB within ten (10) calendar days of learning of the problem. The sponsor-investigator will also report serious, unexpected, suspected adverse reactions and other significant safety information to FDA as required under 21 CFR 312.32.

Adverse events grade 3 and higher, as well as AEs requiring clinical intervention/dose modification, ECIs, and SAEs of any grade, will be reported from the time of signing of consent up until 90 days following the last dose of pembrolizumab.

If a problem, event or information is determined to be an unanticipated problem involving risks to participants or others, it will be reviewed by the convened IRB, appropriate steps will be taken and it will be reported to appropriate institutional and governmental officials as provided under applicable law.

For the purposes of this protocol, the terms Adverse Event, Serious Adverse Event (Related, Possibly Related or Unexpected) and Unanticipated Problem are defined in accordance with the most current Fred Hutchinson Cancer Research Center Institutional Review Board Policy 2.6.

## **Routine Reporting**

Routine reporting is required for all grade 3, 4 and 5 adverse events. Routine reporting will be conducted in accordance with applicable FDA regulations, and agreements with Merck.

#### **Expedited Reporting**

With respect to each research study he or she is conducting, the principal investigator must ensure that the following problems, events, and information involving risks to research participants or others are reported to the IRB not later than ten (10) calendar days after he or she first becomes aware of the problem, event, or information.

## **Adverse Events Requiring Expedited Reporting**

Adverse events require expedited reporting if they meet all three of the following criteria:

- (1) unexpected, and
- (2) related or possibly related to the research and
- (3) serious or suggest that the research places research participants or others at a greater risk of physical or psychological harm than was previously known or recognized.

Unless otherwise specified in the Protocol, therapeutic oncology protocols are not required to specify monitoring parameters for Grade I or II toxicities as described in the Common Terminology Criteria for Adverse Events published by the National Cancer Institute. These adverse events are expected and occur routinely in the subject population being studied. They should be monitored and treated in the practice of routine clinical care.

## 8.0 STATISTICAL ANALYSIS PLAN

## 8.1 Statistical Analysis Plan Summary

This is a single-arm phase II study designed to show a statistically significantly improved overall response rate (ORR) from the fixed benchmark of 25%. This rate is based on early data of efficacy of immune checkpoint modulating antibodies used in treating FL in the relapsed and refractory setting (4). Though representing a lower ORR than has been shown for other first-line therapeutic strategies in iBCL (19) this threshold was chosen with consideration for pembrolizumab's novel mechanism of action compared with standard iBCL treatments and the potential for achieving long-term remissions with low toxicity (20).

## 8.2 Statistical Analysis Plan

We shall use the backbone of a Simon two-stage minimax design for this trial with an additional look to potentially stop for futility based on outcomes observed in two specific histology subgroups (follicular lymphoma, marginal-zone lymphoma). With 33 patients, a Simon two-stage minimax design yields 90% to observe an ORR that is statistically significantly higher (at the one-sided significance level of .05) than the fixed ORR rate of 25% if the assumed-true ORR with the regimen currently proposed is 50%. In the first stage, if we observe 4 or fewer responses among 16 patients (25% or less), consideration will be given to terminating the study due to lack of sufficient efficacy. On the other hand, if 5 or more responses are seen among the first 16 patients (and observed ORR of at least 31%), an additional 17 patients will be enrolled. At this point, if 13 or more responses are seen among the 33 patients (an observed rate of at least 39%), the study will conclude that the proposed treatment is potentially efficacious and worthy of further study.

The modification to the above Simon two-stage design will include an interim look within the first stage, with this interim look consisting of subtype-specific analyses. If there are 0 responses among the first 6 patients with follicular lymphoma, accrual of such patients will be stopped. The same rule will be applied to patients with marginal-zone lymphoma. If the true probability of response is 50%, the probability of seeing 0 responses among 6 patients is .016. This additional look has a small impact on the power of the Simon design (since, under the alternative hypothesis, we may incorrectly stop at least one group for futility, hence decreasing the power (i.e., increasing the Type II error or false negative rate). In particular, if one assumes a 50% ORR (consistent with the alternative hypothesis in the Simon design) in both subtypes with an equal probability of enrollment to each subtype, the addition of the subtype-specific rules from above decreases the power from 90% approximately 87% (estimated from 5,000 simulations). Note that if in each subtype there are 0 responses in the first 6 patients, for a total of 0/12, these results would lead to stopping the trial per the Simon two-stage rules as it would not be possible to achieve at least 5 responses in the first 16 patients.

If the study is stopped due to lack of efficacy in a histologic subgroup, the study may only be reopened to accrual for patients with that histology with modifications (e.g. addition of a

second agent, change in dosing, etc) that have been reviewed and approved where appropriate by the sponsor, scientific review, and relevant regulatory bodies.

## Suspension rules for toxicity:

Prior studies treating patients that have not received prior chemotherapy suggest that the rates of grade ≥3 immune-related AEs occur in approximately 10% of patients (Reck et al, NEJM 2016). Infusion reactions of ≥grade 3 are less common and less consistently reported in publications. For this reason, we will initiate a suspension rule for infusion- or immune-related AEs of ≥grade 3 of up to 12%. This will be deemed to occur if the lower level of a one-sided 80% confidence interval for immune-related or infusional AEs of ≥grade 3 exceeds 12%.

Operationally, the study will be suspended and referred to the DSMC for consideration of results and appropriate modification or termination of the study if

• 3 out of the first 11 or fewer, 5 out of the first 22 or fewer, 6 out of the first 33 or fewer have ≥ grade 3 immune related or infusional AEs

If the true probability of  $\geq$ grade 3 AEs is 5%, the probability of suspending the trial due to excess AEs after 11, 22, and 33 patients is approximately <0.02, 0.02, and 0.02, respectively. If the true probability of  $\geq$ grade 3 AEs is 30%, the probability of suspension due to excess AE is approximately 0.80, 0.94, and 0.99, respectively. (Probabilities of suspension estimated from 5,000 simulations).

## 8.3 Efficacy Analysis

Response assessments will be performed as described in Section 7.1.2.5.

#### 8.3.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the overall response rate (CR + PR for FL and MZL) and will be calculated for all treated patients. The corresponding 95% two-sided confidence interval will be derived.

#### 8.3.2 Secondary Efficacy Endpoints

#### **8.3.2.1** Duration of response

Duration of response will be measured from the time by which the measurement criteria are met for CR or PR, whichever is recorded first, until death or the first date by which recurrent or progressive disease is objectively documented. Subjects who are progression-free and alive at the time of clinical cut-off or have unknown status will be censored at the last tumor assessment.

Non-responders will be excluded from the analysis of DOR. Kaplan Meier methodology will be used to estimate event-free curves.

## 8.3.2.2 Progression-free survival

PFS will be measured for each disease cohort as time from the first study drug administration to the first occurrence of lymphoma progression or death from any cause.

Data for subjects without disease progression or death will be censored at the date of the last tumor assessment. Kaplan-Meier methodology will be used to estimate the event-free curves.

## 8.3.2.3 Time to next therapy

Time to additional anti-neoplastic treatment will be measured from the time of first study drug administration until the date of the first subsequent therapy given to treat the iBCL. Data for subjects that have not received additional anti-neoplastic therapy will be censored at the date of last known contact.

## 8.3.2.4 Safety Analysis

Adverse events and serious adverse events will be reviewed internally on an ongoing basis to identify safety concerns. Safety summaries will include tabulations in the form of tables. The frequency of treatment-emergent AE's will be summarized. Additional AE summaries will include AE frequency by AE severity and relationship to the study drug.

AE's requiring discontinuation of the study drug will be summarized separately, both overall and by AE severity and by relationship to the study drug. Clinically significant abnormal laboratory values will be summarized over study visits.

#### 8.3.2.5 Biomarkers

Biomarker data will be collected on all subjects enrolled on study and examined for correlation of response to pembrolizumab in aggregate and within disease subtypes cohorts. Descriptive statistics will be used for hypothesis-generating endpoints.

## 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

#### 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies will be provided by Merck as summarized in Table 7.

**Table 7 Product Descriptions** 

| Product Name & Potency | Dosage Form |
|------------------------|----------------------------------|
| Pembrolizumab 50 mg | Lyophilized Powder for Injection |

| Product Name & Potency | Dosage Form |
|---------------------------|------------------------|
| Pembrolizumab 100 mg/ 4mL | Solution for Injection |

## 9.2 Packaging and Labeling Information

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

## 9.3 Clinical Supplies Disclosure

This trial is open-label; therefore, the subject, the trial site personnel, the Sponsor-Investigator and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text; random code/disclosure envelopes or lists are not provided.

## 9.4 Storage and Handling Requirements

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

#### 9.5 Returns and Reconciliation

The investigator is responsible for keeping accurate records of the clinical supplies received from Merck or designee, the amount dispensed to and returned by the subjects and the amount remaining at the conclusion of the trial.

Upon completion or termination of the study, all unused and/or partially used investigational product will be destroyed at the site per institutional policy. It is the Investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

## 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

## 10.1 Data and Safety Monitoring Plan

Ongoing trial oversight is carried out by the Principal Investigator and study staff. These individuals will communicate on a regular basis to review recently acquired data and adverse events. The data recorded within the research charts and protocol database is compared with the actual data that is available from the medical record and/or clinical histories. Data detailed

in the research case report forms includes the nature and severity of all toxicities, which are also reported as described above.

Institutional support of trial monitoring will be in accordance with the Fred Hutch/University of Washington Cancer Consortium Institutional Data and Safety Monitoring Plan. Under the provisions of this plan, Fred Hutch Clinical Research Support coordinates data and compliance monitoring conducted by consultants, contract research organizations, or Fred Hutch employees unaffiliated with the conduct of the study. Independent monitoring visits occur at specified intervals determined by the assessed risk level of the study and the findings of previous visits per the institutional DSMP.

In addition, protocols are reviewed at least annually and as needed by the Consortium Data and Safety Monitoring Committee (DSMC), Fred Hutch Scientific Review Committee (SRC) and the Fred Hutch/University of Washington Cancer Consortium Institutional Review Board (IRB). The review committees evaluate accrual, adverse events, stopping rules, and adherence to the applicable data and safety monitoring plan for studies actively enrolling or treating patients. The IRB reviews the study progress and safety information to assess continued acceptability of the risk-benefit ratio for human subjects. Approval of committees as applicable is necessary to continue the study.

The trial will comply with the standard guidelines set forth by these regulatory committees and other institutional, state, and federal guidelines.

#### 10.2 Records

Research staff under the supervision of the investigators will maintain case report forms and secured databases on the relevant clinical and laboratory data. Records maintained in investigators' offices will be secured with access limited to study personnel. Authorization for access to medical records will be obtained from all patients in accordance with provisions of the Health Insurance Portability and Accountability Act (HIPAA).

## 10.3 Regulatory Responsibilities of Sponsor-Investigator

The Sponsor-Investigator will ensure that the study is conducted in accordance with all applicable institutional, state, and federal regulatory requirements, including, but not limited to: compliance with requirements for IRB and other regulatory approvals, monitoring responsibilities, reporting obligations, and compliance with standards for written informed consent from all patients entering the study. In addition, the investigator will ensure oversight of the study via data and safety monitoring as described above.

#### REFERENCES

- 1. Martin P, Chadburn A, Christos P, Weil K, Furman RR, Ruan J, et al. Outcome of deferred initial therapy in mantle-cell lymphoma. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology.* 2009;27(8):1209-13.
- 2. Dave SS, Wright G, Tan B, Rosenwald A, Gascoyne RD, Chan WC, et al. Prediction of survival in follicular lymphoma based on molecular features of tumor-infiltrating immune cells. *The New England journal of medicine*. 2004;351(21):2159-69.
- 3. Berger R, Rotem-Yehudar R, Slama G, Landes S, Kneller A, Leiba M, et al. Phase I safety and pharmacokinetic study of CT-011, a humanized antibody interacting with PD-1, in patients with advanced hematologic malignancies. *Clinical cancer research:* an official journal of the American Association for Cancer Research. 2008;14(10):3044-51.
- 4. Lesokhin AM, Ansell SM, Armand P, Scott EC, Halwani A, Gutierrez M, et al. ASH Conference; 2014:291-.
- 5. Westin JR, Chu F, Zhang M, Fayad LE, Kwak LW, Fowler N, et al. Safety and activity of PD1 blockade by pidilizumab in combination with rituximab in patients with relapsed follicular lymphoma: a single group, open-label, phase 2 trial. *The lancet oncology*. 2014;15(1):69-77.
- 6. Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. *Nature reviews Cancer*. 2012;12(4):252-64.
- 7. Glimelius B, and Lahn M. Window-of-opportunity trials to evaluate clinical activity of new molecular entities in oncology. *Annals of oncology: official journal of the European Society for Medical Oncology / ESMO*. 2011;22(8):1717-25.
- 8. Disis ML. Immune regulation of cancer. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology.* 2010;28(29):4531-8.
- 9. Francisco LM, Sage PT, and Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. *Immunological reviews*. 2010;236:219-42.
- 10. Talmadge JE, Donkor M, and Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. *Cancer metastasis reviews*. 2007;26(3-4):373-400.
- 11. Horning SJ, and Rosenberg SA. The natural history of initially untreated low-grade non-Hodgkin's lymphomas. *The New England journal of medicine*. 1984;311(23):1471-5.
- 12. Drobyski WR, and Qazi R. Spontaneous regression in non-Hodgkin's lymphoma: clinical and pathogenetic considerations. *American journal of hematology*. 1989;31(2):138-41.
- 13. Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, et al. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. *Clinical cancer research: an official journal of the American Association for Cancer Research.* 2014;20(19):5064-74.
- 14. Carbone DP, Socinski MA, Chen AC, Bhagavatheeswaran P, Reck M, and Paz-Ares L. A phase III, randomized, open-label trial of nivolumab (anti-PD-1; BMS-936558, ONO-4538) versus investigator's choice chemotherapy (ICC) as first-line therapy for stage IV or recurrent PD-L1+ non-small cell lung cancer (NSCLC). *ASCO Meeting Abstracts*. 2014;32(15\_suppl):TPS8128.

- 15. Gettinger SN, Shepherd FA, Antonia SJ, Brahmer JR, Chow LQM, Juergens RA, et al. First-line nivolumab (anti-PD-1; BMS-936558, ONO-4538) monotherapy in advanced NSCLC: Safety, efficacy, and correlation of outcomes with PD-L1 status. *ASCO Meeting Abstracts*. 2014;32(15\_suppl):8024.
- 16. Wang Q, Gao J, and Wu X. Pseudoprogression and hyperprogression after checkpoint blockade. *International immunopharmacology*. 2018;58:125-35.
- 17. Champiat S, Dercle L, Ammari S, Massard C, Hollebecque A, Postel-Vinay S, et al. Hyperprogressive Disease Is a New Pattern of Progression in Cancer Patients Treated by Anti-PD-1/PD-L1. Clinical cancer research: an official journal of the American Association for Cancer Research. 2017;23(8):1920-8.
- 18. Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. *Journal of clinical oncology:* official journal of the American Society of Clinical Oncology. 2014;32(27):3059-68.
- 19. Kahl BS, Hong F, Williams ME, Gascoyne RD, Wagner LI, Krauss JC, et al. Rituximab extended schedule or re-treatment trial for low-tumor burden follicular lymphoma: eastern cooperative oncology group protocol e4402. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology.* 2014;32(28):3096-102.
- 20. Moreno BH, and Ribas A. Anti-programmed cell death protein-1/ligand-1 therapy in different cancers. *British journal of cancer*. 2015.
- 21. Solal-Céligny P, Roy P, Colombat P, White J, Armitage JO, Arranz-Saez R, et al. Follicular lymphoma international prognostic index. *Blood.* 2004;104(5):1258-65.

#### 11.0 APPENDICES

## 11.1 ECOG Performance Status

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |

<sup>\*</sup> As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982. The Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.

## 11.2 Common Terminology Criteria for Adverse Events V4.0 (CTCAE)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

## 11.3 Response Evaluation

## 11.3.1 The Lugano Response Classification: For FL and MZL (18)

| Response and<br>Site | PET-CT-Based Response | CT-Based Response |
|---|---|---|
| Complete | Complete metabolic response | Complete radiologic response (all of the following) |
| | Score 1, 2, or $3^*$ with or without a residual mass on $5PS^{\dagger}$ | Target nodes/nodal masses must regress to ≤ 1.5 cm in LDi |
| | It is recognized that in Waldeyer's ring or extranodal<br>sites with high physiologic uptake or with activation<br>within spleen or marrow (eg, with chemotherapy or<br>myeloid colony-stimulating factors), uptake may be | |
| Lymph nodes and | greater than normal mediastinum and/or liver. In this | |
| extralymphatic | circumstance, complete metabolic response may be | |
| sites | inferred if uptake at sites of initial involvement is no | No extralymphatic sites of disease |

| Response and<br>Site | PET-CT-Based Response | CT-Based Response |
|---|---|---|
| | greater than surrounding normal tissue even if the tissue has high physiologic uptake | |
| Nonmeasured lesion | Not applicable | Absent |
| Organ enlargement | Not applicable | Regress to normal |
| New lesions | None | None |
| Bone marrow | No evidence of FDG-avid disease in marrow | Normal by morphology; if indeterminate, IHC negative |
| Partial | Partial metabolic response | Partial remission (all of the following) |
| Lymph<br>nodes and<br>extralymphatic<br>sites | Score 4 or 5† with reduced uptake compared with baseline and residual mass(es) of any size | ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites |
| | At interim, these findings suggest responding disease | When a lesion is too small to measure on CT, assign 5 mm × 5 mm as the default value |
| | At end of treatment, these findings indicate residual disease | When no longer visible, $0 \times 0$ mm |
| | | For a node > 5 mm × 5 mm, but smaller than normal, use actual measurement for calculation |
| Nonmeasured lesions | Not applicable | Absent/normal, regressed, but no increase |
| Organ enlargement | Not applicable | Spleen must have regressed by > 50% in length beyond normal |
| New lesions | None | None |
| | Residual uptake higher than uptake in normal marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). If there are persistent focal changes in the marrow in the context of a nodal response, consideration should be given to further evaluation with | |
| Bone marrow | MRI or biopsy or an interval scan | Not applicable |
| No response or stable disease | No metabolic response | Stable disease |
| Target<br>nodes/nodal<br>masses,<br>extranodal lesions | Score 4 or 5 with no significant change in FDG uptake from baseline at interim or end of treatment | < 50% decrease from baseline in SPD<br>of up to 6 dominant, measurable nodes<br>and extranodal sites; no criteria for<br>progressive disease are met |

| Response and | DETECT D. LD. | CT D I D |
|---|---|---|
| Site | PET-CT-Based Response | CT-Based Response |
| Nonmeasured lesions | Not applicable | No increase consistent with progression |
| Organ<br>enlargement | Not applicable | No increase consistent with progression |
| New lesions | None | None |
| Bone marrow | No change from baseline | Not applicable |
| Progressive disease | Progressive metabolic disease | Progressive disease requires at least 1 of the following |
| Individual target nodes/nodal masses Extranodal lesions | Score 4 or 5 with an increase in intensity of uptake from baseline and/or New FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment | PPD progression: An individual node/lesion must be abnormal with: LDi > 1.5 cm and Increase by $\geq 50\%$ from PPD nadir and An increase in LDi or SDi from nadir 0.5 cm for lesions $\leq 2$ cm 1.0 cm for lesions $\geq 2$ cm In the setting of splenomegaly, the splenic length must increase by $\geq 50\%$ of the extent of its prior increase beyond baseline (eg, a 15-cm spleen must increase to $\geq 16$ cm). If no prior splenomegaly, must increase by at least 2 cm from baseline New or recurrent splenomegaly |
| Nonmeasured<br>lesions | None | New or clear progression of preexisting nonmeasured lesions |
| New lesions | New FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation). If uncertain regarding etiology of new lesions, biopsy or interval scan may be considered | Regrowth of previously resolved lesions A new node > 1.5 cm in any axis A new extranodal site > 1.0 cm in any axis; if < 1.0 cm in any axis, its presence must be unequivocal and must be attributable to lymphoma Assessable disease of any size unequivocally attributable to lymphoma |
| Bone marrow | New or recurrent FDG-avid foci | New or recurrent involvement |

- Abbreviations: 5PS, 5-point scale; CT, computed tomography; FDG, fluorodeoxyglucose; IHC, immunohistochemistry; LDi, longest transverse diameter of a lesion; MRI, magnetic resonance imaging; PET, positron emission tomography; PPD, cross product of the LDi and perpendicular diameter; SDi, shortest axis perpendicular to the LDi; SPD, sum of the product of the perpendicular diameters for multiple lesions.
- A score of 3 in many patients indicates a good prognosis with standard treatment, especially if at the time of an interim scan. However, in trials involving PET where deescalation is investigated, it may be preferable to consider a score of 3 as inadequate response (to avoid undertreatment). Measured dominant lesions: Up to six of the largest dominant nodes, nodal masses, and extranodal lesions selected to be clearly measurable in two diameters. Nodes should preferably be from disparate regions of the body and should include, where applicable, mediastinal and retroperitoneal areas. Non-nodal lesions include those in solid organs (eg, liver, spleen, kidneys, lungs), GI involvement, cutaneous lesions, or those noted on palpation. Nonmeasured lesions: Any disease not selected as measured, dominant disease and truly assessable disease should be considered not measured. These sites include any nodes, nodal masses, and extranodal sites not selected as dominant or measurable or that do not meet the requirements for measurability but are still considered abnormal, as well as truly assessable disease, which is any site of suspected disease that would be difficult to follow quantitatively with measurement, including pleural effusions, ascites, bone lesions, leptomeningeal disease, abdominal masses, and other lesions that cannot be confirmed and followed by imaging. In Waldeyer's ring or in extranodal sites (eg, GI tract, liver, bone marrow), FDG uptake may be greater than in the mediastinum with complete metabolic response, but should be no higher than surrounding normal physiologic uptake (eg, with marrow activation as a result of chemotherapy or myeloid growth factors).

† PET 5PS: 1, no uptake above background; 2, uptake  $\leq$  mediastinum; 3, uptake > mediastinum but  $\leq$  liver; 4, uptake moderately > liver; 5, uptake markedly higher than

## 11.4 FLIPI Scoring System (21)

Patients diagnosed with FL are assigned points according to the following system; the sum of the points constitutes the FLIPI score:

- 1. Age greater than 60 years
- 2. Stage III or IV disease
- 3. Greater than 4 lymph node groups involved
- 4. Serum hemoglobin less than 12 g/dL
- 5. Elevated serum LDH

#### 11.5 Events of Clinical Interest Guidance Document: Version 5

#### 11.9.1 OVERVIEW

The purpose of this appendix is to provide study sites with guidance on the identification and management of Events of Clinical Interest for the MK-3475 (also known as pembrolizumab) program.

Based on literature review, and consideration of mechanism of action of pembrolizumab, potential immune-related adverse events (irAEs) are the primary Event of Clinical Interest (ECI). Immune-related AEs are adverse events associated with the treatment of patients with immunotherapy treatments that appear to be associated with the immune therapy's mechanism of action. Based on these potential irAEs, the sponsor has defined a list of specific adverse event terms (ECIs) that are selected adverse experiences that must be reported to Merck within 2 business days from the time the Investigator/physician is aware of such an occurrence, regardless of whether or not the investigator/physician considers the event to be related to study drug(s). In addition, these ECIs require additional detailed information to be collected and entered in the study database. ECIs may be identified through spontaneous patient report and/or upon review of subject data. Table 1 provides the list of terms and reporting requirements for AEs that must be reported as ECIs for MK-3475 protocols. Of note, the requirement for reporting of ECIs applies to all arms, including comparators, of MK-3475 clinical trials

Given that our current list of events of clinical interest is not comprehensive for all potential immune-related events, it is possible that AEs other than those listed in this document may be observed in patients receiving pembrolizumab. Therefore, any Grade 3 or higher event that the investigator/physician considers to be immune-related should be reported as an ECI regardless of whether the specific event term is in Table 1 and reported to Merck within 2 business days from the time the Investigator/physician is aware of such an occurrence. Adverse events that are both an SAE and an ECI should be reported one time as an SAE only, however the event must be appropriately identified as an ECI as well in in the database.

**Table 1: Events of Clinical Interest** 

| Pneumonitis (reported as ECI if ≥ Grade 2) | | |
|---|---|---|
| Acute interstitial pneumonitis | Interstitial lung disease | Pneumonitis |
| Colitis (reported as ECI if ≥ Grade 2 | or any grade resulting in dose modific | cation or use of systemic steroids to treat |
| Intestinal Obstruction | Colitis | Colitis microscopic |
| Enterocolitis | Enterocolitis hemorrhagic | Gastrointestinal perforation |
| Necrotizing colitis | Diarrhea | |
| Endocrine (reported as ECI if $\geq$ Grade 3 or $\geq$ Grade 2 and resulting in dose modification or use of systemic | | |
| steroids to treat the AE) | | |
| Adrenal Insufficiency | Hyperthyroidism | Hypophysitis |
| Hypopituitarism | Hypothyroidism | Thyroid disorder |
| Thyroiditis | Hyperglycemia, if ≥Grade 3 and associated with ketosis or metabolic acidosis | |
| Endocrine (reported as ECI) | | |
| Type 1 diabetes mellitus (if new onset) | | |

| Hematologic (reported as ECI if $\geq$ Grade 3 or any grade resulting in dose modification or use of systemic steroids to treat the AE) | | |
|---|---|---|
| Autoimmune hemolytic anemia | Aplastic anemia | Thrombotic Thrombocytopenic Purpura (TTP) |
| Idiopathic (or immune) Thrombocytopenia Purpura (ITP) Any Grade 4 anemia regardless of under | Disseminated Intravascular Coagulation (DIC) | Haemolytic Uraemic Syndrome (HUS) |
| , | , <u> </u> | ation or use of systemic steroids to treat the |
| Hepatitis | Autoimmune hepatitis | Transaminase elevations (ALT and/o |
| Infusion Reactions (reported as ECI f | • | |
| Allergic reaction | Anaphylaxis | Cytokine release syndrome |
| Serum sickness | Infusion reactions | Infusion-like reactions |
| Neurologic (reported as ECI for any g | rade) | |
| Autoimmune neuropathy | Guillain-Barre syndrome | Demyelinating polyneuropathy |
| Myasthenic syndrome | | |
| Ocular (report as ECI if ≥ Grade 2 or | any grade resulting in dose modificati | on or use of systemic steroids to treat the |
| Uveitis | Iritis | |
| Renal (reported as ECI if $\geq$ Grade 2) | | |
| Nephritis | Nephritis autoimmune | Renal Failure |
| Renal failure acute Creatinine elevations (report as ECI if \(\geq\)Grade 3 or any grade resulting in doso modification or use of systemic steroids to treat the AE) | | |
| Skin (reported as ECI for any grade) | | |
| Dermatitis exfoliative | Erythema multiforme | Stevens-Johnson syndrome |
| Toxic epidermal necrolysis | | |
| Skin (reported as ECI if ≥ Grade 3) | | |
| Pruritus | Rash | Rash generalized |
| Rash maculo-papular | | |
| Any rash considered clinically significant in the physician's judgment | | |
| Other (reported as ECI for any grade) | | |
| Myocarditis Pancreatitis Pericarditis | | Pericarditis |
| Any other Grade 3 event which is consider | ered immune-related by the physician | |

Each of the events above is described within this guidance document, along with site requirements for reporting these events to the Sponsor. The information collected should be entered into the narrative field(s) of the Adverse Event module in the database (please note, if narrative entry into the database is not available, please use the narrative text box on the 1727/AER Form). If additional Medical History or Concomitant Medications are reported, the Medical History and Concomitant Medication modules in the database must be updated.

In addition, the guidelines include recommendations on the management of these ECIs. These guidelines are intended to be applied when the physician determines the events to be related to pembrolizumab. Note: if after the evaluation the event is determined not to be related, the physician is instructed to follow the ECI reporting guidance but does not need to follow the treatment guidance (below). Therefore, these recommendations should be seen as guidelines and the treating physician should exercise individual clinical judgment based on the patient. For any question of dose modification or other treatment options, the specific language in the

protocol should be followed. Any questions pertaining to the collection of this information or management of ECIs should be directed to your local Sponsor contact.

#### **Dose Modification/Discontinuation**

The treatment guidance provides specific direction when to hold and/or discontinue pembrolizumab for each immune related adverse event. Of note, when the guidance states to "discontinue" pembrolizumab this is the permanent discontinuation of treatment with pembrolizumab. "Hold" means to stop treating with pembrolizumab but resumption of treatment may be considered assuming the patient meets the criteria for resumption of treatment.

#### 2. ECI REPORTING GUIDELINES

ECIs are selected non-serious and serious adverse experiences that must be reported to Merck within 2 business days regardless of attribution to study treatment. The AEs listed in this document and any event that meets the ECI criteria (as noted) in Table 1 or in the respective protocol (event term and Grade) must be reported regardless of physician-determined causality with study medication and whether or not considered immune-related by the physician (unless otherwise specified).

Physicians/study coordinators/designated site personnel are required to record these experiences as ECIs on the Adverse Experience electronic Case Report Forms (eCRFs) (or on paper) and to provide supplemental information (such as medical history, concomitant medications, investigations, etc.) about the event.

- Please refer to the Data Entry Guidelines (DEGs) for your protocol.
- Please refer to protocol for details on reporting timelines and reporting of Overdose and Drug Induced Liver Injury (DILI).

#### 3. ECI CATEGORIES AND TERMS

This section describes the ECI categories and outlines subject management guidelines when an ECI is reported.

#### 3.1 Pneumonitis

The following AE terms, if considered ≥ Grade 2, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Pneumonitis
- Interstitial lung disease

Acute interstitial pneumonitis

If symptoms indicate possible new or worsening cardiac abnormalities additional testing and/or a cardiology consultation should be considered.

All attempts should be made to rule out other causes such as metastatic disease, bacterial or viral infection. It is important that patients with a suspected diagnosis of pneumonitis be managed as per the guidance below until treatment-related pneumonitis is excluded. Treatment of both a potential infectious etiology and pneumonitis in parallel may be warranted. Management of the treatment of suspected pneumonitis with steroid treatment should not be delayed for a therapeutic trial of antibiotics. If an alternative diagnosis is established, the patient does not require management as below; however the AE should be reported regardless of etiology.

#### **Course of Action**

#### Grade 2 events:

- Report as ECI
- Hold pembrolizumab.
- Consider pulmonary consultation with bronchoscopy and biopsy/BAL.
- Consider ID consult
- Conduct an in-person evaluation approximately twice per week
- Consider frequent Chest X-ray as part of monitoring
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg/day prednisone or equivalent. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- Second episode of pneumonitis discontinue pembrolizumab if upon re-challenge the patient develops a second episode of Grade 2 or higher pneumonitis.

#### Grade 3 and 4 events:

- Report as ECI
- Discontinue pembrolizumab.
- Hospitalize patient
- Bronchoscopy with biopsy and/or BAL is recommended.
- Immediately treat with intravenous steroids (methylprednisolone 125 mg IV). When symptoms improve to Grade 1 or less, a high dose oral steroid (prednisone 1 to 2 mg/kg once per day or dexamethasone 4 mg every 4 hours) taper should be started and continued over no less than 4 weeks.
- If IV steroids followed by high dose oral steroids does not reduce initial symptoms within 48 to 72 hours, treat with additional anti-inflammatory measures. Discontinue additional anti-inflammatory measures upon symptom relief and initiate a prolonged steroid taper over 45 to 60 days. If symptoms worsen during steroid reduction, initiate a retapering of steroids starting at a higher dose of 80 or 100 mg followed by a more prolonged taper and administer additional anti-inflammatory measures, as

needed

Add prophylactic antibiotics for opportunistic infections.

#### 3.2 Colitis

The following AE terms, if considered  $\geq$  Grade 2 or resulting in dose modification or use of systemic steroids to treat the AE, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Colitis
- Colitis microscopic
- Enterocolitis
- Enterocolitis hemorrhagic
- Gastrointestinal perforation
- Intestinal obstruction
- Necrotizing colitis
- Diarrhea

All attempts should be made to rule out other causes such as metastatic disease, bacterial or parasitic infection, viral gastroenteritis, or the first manifestation of an inflammatory bowel disease by examination for stool leukocytes, stool cultures, a Clostridium difficile titer and endoscopy. However, the AE should be reported regardless of etiology.

#### **Course of Action**

Grade 2 Diarrhea/Colitis (4-6 stools/day over baseline, dehydration requiring IV fluids < 2 business days, abdominal pain, mucus or blood in stool):

- Report as ECI
- Hold pembrolizumab.
- Symptomatic Treatment
- For Grade 2 diarrhea that persists for greater than 3 days, and for diarrhea with blood and/or mucus,
- Consider GI consultation and endoscopy to confirm or rule out colitis
- Administer oral corticosteroids (prednisone 1-2 mg/kg QD or equivalent)
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- If symptoms worsen or persist > 3 days treat as Grade 3

Grade 3 Diarrhea/Colitis (or Grade 2 diarrhea that persists for > 1 week):

Report as ECI

- Hold pembrolizumab.
- Rule out bowel perforation. Imaging with plain films or CT can be useful.
- Recommend consultation with Gastroenterologist and confirmation biopsy with endoscopy.
- Treat with intravenous steroids (methylprednisolone 125 mg) followed by high dose oral steroids (prednisone 1 to 2 mg/kg once per day or dexamethasone 4 mg every 4 hours) When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Taper over 6 to 8 weeks in patients with diffuse and severe ulceration and/or bleeding.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- If IV steroids followed by high dose oral steroids does not reduce initial symptoms within 48 to 72 hours, consider treatment with additional anti-inflammatory measures as described in the literature [5]. Discontinue additional anti-inflammatory measures upon symptom relief and initiate a prolonged steroid taper over 45 to 60 days. If symptoms worsen during steroid reduction, initiate a retapering of steroids starting at a higher dose of 80 or 100 mg followed by a more prolonged taper and administer additional anti-inflammatory measures as needed.

#### Grade 4 events:

- Report as ECI
- Permanently discontinue pembrolizumab.
- Manage as per Grade 3.

## 3.3 Endocrine

The following AE terms, if considered ≥Grade 3 or if ≥Grade 2 and require holding/discontinuation/ modification of pembrolizumab dosing, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Adrenal insufficiency
- Hyperthyroidism
- Hypophysitis
- Hypopituitarism
- Hypothyroidism
- Thyroid disorder
- Thyroiditis

All attempts should be made to rule out other causes such as brain metastases, sepsis and/or infection. However, the AE should be reported regardless of etiology.

## Hypophysitis or other symptomatic endocrinopathy other than hypo- or

#### <u>hvperthvroidism</u>

Grade 2-4 events:

- Report as ECI if appropriate
- Hold pembrolizumab
- Rule out infection and sepsis with appropriate cultures and imaging.
- Monitor thyroid function or other hormonal level tests and serum chemistries more frequently until returned to baseline values.
- Pituitary gland imaging should be considered (MRIs with gadolinium and selective cuts of the pituitary can show enlargement or heterogeneity and confirm the diagnosis).
- Treat with prednisone 40 mg p.o. or equivalent per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- Hypophysitis with clinically significant adrenal insufficiency and hypotension, dehydration, and electrolyte abnormalities (such as hyponatremia and hyperkalemia) constitutes adrenal crisis.
- Consultation with an endocrinologist may be considered.

## **Hyperthyroidism and Hypothyroidism**

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.

Grade 2 hyperthyroidism, Grade 2-4 hypothyroidism events:

- Report as ECI if appropriate (see Table 1)
- Monitor thyroid function or other hormonal level tests and serum chemistries more frequently until returned to baseline values.
- Thyroid hormone and/or steroid replacement therapy to manage adrenal insufficiency.
- Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted.
- In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
- In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- Consultation with an endocrinologist may be considered.

## Grade 3 hyperthyroidism events:

- Report as ECI
- Hold pembrolizumab.
- Rule out infection and sepsis with appropriate cultures and imaging.
- Treat with an initial dose of methylprednisolone 1 to 2 mg/kg intravenously followed by oral prednisone 1 to 2 mg/kg per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 4 hyperthyroidism events:

- Report as ECI
- Discontinue pembrolizumab.
- Manage as per Grade 3

## Type 1 diabetes mellitus (if new onset) and ≥ Grade 3 Hyperglycemia

The following AE terms are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Type I diabetes mellitus (T1DM), if new onset, including diabetic ketoacidosis (DKA)
- Grade 3 or higher hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA).

Immune-mediated diabetes may present as new onset of Type 1 diabetes or an abrupt worsening of pre- existing diabetes associated with laboratorial evidence of beta cell failure. All attempts should be made to rule out other causes such as type 2 diabetes mellitus (T2DM), T2DM decompensation, steroid-induced diabetes, physiologic stress-induced diabetes, or poorly controlled pre-existing diabetes (either T1DM or T2DM), but events meeting the above criteria should be reported as ECIs regardless of etiology. The patients may present with hyperglycemia (abrupt onset or abrupt decompensation) with clinical evidence of diabetic ketoacidosis or laboratory evidence of insulin deficiency, such as ketonuria, laboratory evidence of metabolic acidosis, or low or undetected c-peptide.

#### **Course of Action**

#### T1DM should be immediately treated with insulin.

T1DM or Grade 3-4 Hyperglycemia events:

- Report as ECI if appropriate (see Table 1)
- Hold pembrolizumab for new onset Type 1 diabetes mellitus or Grade 3-4 hyperglycemia associated with evidence of beta cell failure, and resume pembrolizumab when patients are clinically and metabolically stable.
- Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
- Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.
- Consultation with an Endocrinologist is recommended.
- Consider local testing for islet cell antibodies and antibodies to GAD, IA-2, ZnT8, and insulin may be obtained.

## 3.4 Hematologic

The following AE term, if considered Grade  $\geq 3$  or requiring dose modification or use of systemic steroids to treat the AE, are considered an ECI and should be reported to the Sponsor within 2 business days of the event:

- Autoimmune hemolytic anemia
- Aplastic anemia
- Disseminated Intravascular Coagulation (DIC)
- Haemolytic Uraemic Syndrome (HUS)
- Idiopathic (or immune) Thrombocytopenia Purpura (ITP)
- Thrombotic Thrombocytopenic Purpura (TTP)
- Any Grade 4 anemia regardless of underlying mechanism

All attempts should be made to rule out other causes such as metastases, sepsis and/or infection. Relevant diagnostic studies such as peripheral blood smear, reticulocyte count, LDH, haptoglobin, bone marrow biopsy or Coomb's test, etc., should be considered to confirm the diagnosis. However, the AE should be reported regardless of etiology.

#### **Course of Action**

Grade 2 events:

- Report as ECI
- Hold pembrolizumab
- Prednisone 1-2 mg/kg daily may be indicated
- Consider Hematology consultation.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 3 events:

- Report as ECI
- Hematology consultation.
- Hold pembrolizumab Discontinuation should be considered as per specific protocol guidance.
- Treat with methylprednisolone 125 mg iv or prednisone 1-2 mg/kg p.o. (or equivalent) as appropriate
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 4 events:

- Report as ECI
- Hematology consultation
- Discontinue pembrolizumab for all solid tumor indications; refer to protocol for hematologic malignancies.
- Treat with methylprednisolone 125 mg iv or prednisone 1-2 mg/kg p.o. (or equivalent) as appropriate

## 3.5 Hepatic

The following AE terms, if considered  $\geq$  Grade 2 or greater (or any grade with dose modification or use of systemic steroids to treat the AE), are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Autoimmune hepatitis
- Hepatitis
- Transaminase elevations

All attempts should be made to rule out other causes such as metastatic disease, infection or other hepatic diseases. However, the AE should be reported regardless of etiology.

#### Drug Induced Liver Injury (DILI)

In addition, the event must be reported as a Drug Induced Liver Injury (DILI) ECI, if the patient meets the laboratory criteria for potential DILI defined as:

- An elevated alanine transaminase (ALT) or aspartate transaminase (AST) lab value that is greater than or equal to three times (3X) the upper limit of normal (ULN) and
- An elevated total bilirubin lab value that is greater than or equal to two times (2X) ULN and
- At the same time, an alkaline phosphatase (ALP) lab value that is less than 2X ULN,
- As a result of within-protocol-specific testing or unscheduled testing.

Note that any hepatic immune ECI meeting DILI criteria should only be reported once as a DILI event.

#### **Course of Action**

#### Grade 2 events:

- Report as ECI
- Hold pembrolizumab when AST or ALT >3.0 to 5.0 times ULN and/or total bilirubin >1.5 to 3.0 times ULN. In the case of Gilbert's syndrome where baseline bilirubin > 1.5 ULN, hold pembrolizumab when bilirubin > 1.5 to 3.0 times baseline level
- Monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with 0.5-1 mg/kg/day methylprednisolone or oral equivalent and when LFT returns to grade 1 or baseline, taper steroids over at least 1 month, consider prophylactic antibiotics for opportunistic infections, and resume pembrolizumab per protocol
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- Permanently discontinue pembrolizumab for patients with liver metastasis who begin treatment with Grade 2 elevation of AST or ALT, and AST or ALT increases ≥50% relative to baseline and lasts ≥1 week.

## Grade 3 events:

- Report as ECI
- Discontinue pembrolizumab when AST or ALT >5.0 times ULN and/or total bilirubin >3.0 times ULN.
- Consider appropriate consultation and liver biopsy to establish etiology of hepatic injury, if necessary
- Treat with high-dose intravenous glucocorticosteroids for 24 to 48 hours. When symptoms improve to Grade 1 or less, a steroid taper with dexamethasone 4 mg every 4 hours or prednisone at 1 to 2 mg/kg should be started and continued over no less than 4 weeks.
- If serum transaminase levels do not decrease 48 hours after initiation of systemic steroids, oral mycophenolate mofetil 500 mg every 12 hours may be given.
   Infliximab is not recommended due to its potential for hepatotoxicity.
- Several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 4 events:

Report as ECI

- Permanently discontinue pembrolizumab
- Manage patient as per Grade 3 above

## 3.6 Neurologic

The following AE terms, regardless of grade, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Autoimmune neuropathy
- Demyelinating polyneuropathy
- Guillain-Barre syndrome
- Myasthenic syndrome

All attempts should be made to rule out other causes such as metastatic disease, other medications or infectious causes. However, the AE should be reported regardless of etiology.

#### **Course of Action**

#### Grade 2 events:

- Report as ECI
- Moderate (Grade 2) consider withholding pembrolizumab.
- Consider treatment with prednisone 1-2 mg/kg p.o. daily as appropriate
- Consider Neurology consultation. Consider biopsy for confirmation of diagnosis.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 3 and 4 events:

- Report as ECI
- Discontinue pembrolizumab
- Obtain neurology consultation. Consider biopsy for confirmation of diagnosis
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day. If condition worsens consider IVIG or other immunosuppressive therapies as per local guidelines

When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

#### 3.7 Ocular

The following AE terms, if considered Grade ≥2 or requiring dose modification or use of systemic steroids to treat the AE, is considered an ECI and should be reported to the Sponsor within 2 business days of the event:

Uveitis

- Iritis

All attempts should be made to rule out other causes such as metastatic disease, infection or other ocular disease (e.g. glaucoma or cataracts). However, the AE should be reported regardless of etiology.

#### **Course of Action**

#### Grade 2 events:

- Evaluation by an ophthalmologist is strongly recommended.
- Treat with topical steroids such as 1% prednisolone acetate suspension and iridocyclitics.
- Discontinue pembrolizumab as per protocol if symptoms persist despite treatment with topical immunosuppressive therapy.

#### Grade 3 events:

- Evaluation by an ophthalmologist is strongly recommended
- Hold pembrolizumab and consider permanent discontinuation as per specific protocol guidance.
- Treat with systemic corticosteroids such as prednisone at a dose of 1 to 2 mg/kg per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 4 events:

- Evaluation by an ophthalmologist is strongly recommended
- Permanently discontinue pembrolizumab.
- Treat with corticosteroids as per Grade 3 above

#### 3.8 Renal

The following AEs if  $\geq$  Grade 2 are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Nephritis
- Nephritis autoimmune
- Renal failure
- Renal failure acute

Creatinine elevations  $\geq$  Grade 3 or any grade with dose modification or use of systemic steroids to treat the AE.

All attempts should be made to rule out other causes such as obstructive uropathy, progression of disease, or injury due to other chemotherapy agents. A renal consultation is recommended. However, the AE should be reported regardless of etiology.

#### **Course of Action**

#### Grade 2 events:

- Hold pembrolizumab
- Treatment with prednisone 1-2 mg/kg p.o. daily.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 3-4 events:

- Discontinue pembrolizumab
- Renal consultation with consideration of ultrasound and/or biopsy as appropriate
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone IV or equivalent once per day.

When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

## 3.9 Skin

## Rash and Pruritus

The following AEs should be considered as ECIs, if  $\geq$  Grade 3 and should be reported to the Sponsor within 2 business days of the event:

- Pruritus
- Rash
- Rash generalized
- Rash maculo-papular
- In addition to CTCAE Grade 3 rash, any rash that is considered clinically significant, in the physician's judgment, should be treated as an ECI. Clinical significance is left to the physician to determine, and could possibly include rashes

- such as the following:
- rash with a duration >2 weeks; OR
- rash that is >10% body surface area; OR
- rash that causes significant discomfort not relieved by topical medication or temporary cessation of study drug.

#### Other Skin ECIs

The following AEs should **always** be reported as ECIs, regardless of grade, and should be reported to the Sponsor within 2 business days of the event:

- Dermatitis exfoliative
- Erythema multiforme
- Steven's Johnson syndrome
- Toxic epidermal necrolysis

Please note, the AE should be reported regardless of etiology.

#### **Course of Action**

Grade 2 events:

- Symptomatic treatment should be given such as topical glucocorticosteroids (e.g., betamethasone 0.1% cream or hydrocortisone 1%) or urea-containing creams in combination with oral anti-pruritics (e.g., diphenhydramine HCl or hydroxyzine HCl).
- Treatment with oral steroids is at physician's discretion for Grade 2 events.

#### Grade 3 events:

- Hold pembrolizumab.
- Consider Dermatology Consultation and biopsy for confirmation of diagnosis.
- Treatment with oral steroids is recommended, starting with 1 mg/kg prednisone or equivalent once per day or dexamethasone 4 mg four times orally daily. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 4 events:

- Permanently discontinue pembrolizumab.
- Dermatology consultation and consideration of biopsy and clinical dermatology photograph.
- Initiate steroids at 1 to 2 mg/kg prednisone or equivalent. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

## 3.10 Immediate Evaluation for Potential Skin ECIs

## A. Photographs:

Every attempt should be made to get a photograph of the actual ECI skin lesion or rash as soon as possible. Obtain appropriate consent for subject photographs if a consent form addendum is required by your IRB/ERC.

- Take digital photographs of:
  - o the head (to assess mucosal or eye involvement),
  - o the trunk and extremities, and
  - o a close-up of the skin lesion/rash.
- If possible, a ruler should be placed alongside the site of a skin occurrence as a fixed marker of distance.
- The time/date stamp should be set in the 'ON' position for documentation purposes.
- Photographs should be stored with the subject's study records.
- The Sponsor may request copies of photographs. The local study contact (e.g., CRA) will provide guidance to the site, if needed.

#### **B. Past Medical History**:

Collect past medical history relevant to the event, using the questions in Appendix 2 (Past Medical History Related to Dermatologic Event) as a guide. Any preexisting conditions not previously reported (e.g., drug allergy) should be entered into the Medical History eCRF.

#### C. Presentation of the Event:

Collect information on clinical presentation and potential contributing factors using the questions in Appendix 3 (Presentation of the Dermatologic Event) as a guide. This information should be summarized and entered in narrative format in the AE eCRF. Please use the available free-text fields, such as Signs and Symptoms. Note pertinent negatives where applicable to reflect that the information was collected. Any treatments administered should be entered on the Concomitant Medication eCRF.

## D. Vitals Signs and Standard Laboratory Tests:

Measure vital signs (pulse, sitting BP, oral temperature, and respiratory rate) and record on the Vital Signs eCRF. Perform standard laboratory tests (CBC with manual differential and serum chemistry panel, including LFTs).

#### E. Focused Skin Examination:

Perform a focused skin examination using the questions in Appendix 4 (Focused Skin Examination) as a guide. Information should be summarized and entered on the Adverse Experience eCRF as part of the narrative.

#### F. Dermatology Consult

Refer the subject to a dermatologist as soon as possible.

- For a "severe rash", the subject must be seen within 1-2 days of reporting the event.
- For clinically significant rash, the subject should be seen within 3-5 days.

The dermatologist should submit a biopsy sample to a certified dermatopathology laboratory or to a pathologist experienced in reviewing skin specimens.

The site should provide the dermatologist with all relevant case history, including copies of clinical photographs and laboratory test results.

## 3.11 Other

The following AEs, regardless of grade, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Myocarditis
- Pericarditis
- Pancreatitis
- Any additional Grade 3 or higher event which the physician considers to be immune related

All attempts should be made to rule out other causes. Therapeutic specialists should be consulted as appropriate. However, the AE should be reported regardless of etiology.

#### **Course of Action**

Grade 2 events or Grade 1 events that do not improve with symptomatic treatment:

- Withhold pembrolizumab.
- Systemic corticosteroids may be indicated.
- Consider biopsy for confirmation of diagnosis.
- If pembrolizumab held and corticosteroid required, manage as per grade 3 below.

#### Grade 3 events:

- Hold pembrolizumab
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day.
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks. Otherwise, pembrolizumab treatment may be restarted and the dose modified as specified in the protocol

## Grade 4 events:

- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day. Discontinue pembrolizumab

## 3.12 Infusion Reactions

The following AE terms, regardless of grade, are considered ECIs and should be reported to the Sponsor within 2 business days of the event:

- Allergic reaction
- Anaphylaxis
- Cytokine release syndrome
- Serum sickness
- Infusion reactions
- Infusion-like reactions

## **Course of Action**

Refer to infusion reaction table in the protocol and below.

| NCI CTCAE Grade | Treatment | Premedication at<br>Subsequent Dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |

| Grade 2 | Stop Infusion. | Subject may be premedicated 1.5h |
|---|---|---|
| Requires infusion interruption | Additional appropriate medical therapy may | (± 30 minutes) prior to infusion of |
| but responds promptly to | include but is not limited to: | pembrolizumab with: |
| symptomatic treatment (e.g., | IV fluids Antihistamines NSAIDS | |
| antihistamines, NSAIDS, | Acetaminophen Narcotics | Diphenhydramine 50 mg p.o. (or |
| narcotics, IV fluids); | Increase monitoring of vital signs as medically | equivalent dose of antihistamine). |
| prophylactic medications | indicated until the subject is deemed medically | , |
| indicated for < =24 hrs | stable in the opinion of the investigator. | Acetaminophen 500-1000 mg p.o. |
| | If symptoms resolve within one hour of stopping | (or equivalent dose of antipyretic). |
| | drug infusion, the infusion may be restarted at 50% | |
| | of the original infusion rate (e.g. from 100 mL/hr to | |
| | 50 mL/hr). | |
| | Otherwise dosing will be held until symptoms | |
| | resolve and the subject should be premedicated for | |
| | the next scheduled dose. | |
| | Subjects who develop Grade 2 toxicity despite | |
| | adequate premedication should be permanently | |
| | discontinued from further trial treatment | |
| | administration. | |
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| Grade 3: | Additional appropriate medical therapy may include | |
| Prolonged (i.e., not rapidly | but is not limited to: | |
| responsive to symptomatic | IV fluids Antihistamines NSAIDS | |
| medication and/or brief | Acetaminophen Narcotics | |
| interruption of infusion); | Oxygen Pressors | |
| recurrence of symptoms | Corticosteroids | |
| following initial improvement; | Epinephrine | |
| hospitalization indicated for | | |
| other clinical sequelae (e.g., | Increase monitoring of vital signs as medically | |
| renal impairment, pulmonary | indicated until the subject is deemed medically | |
| infiltrates) | stable in the opinion of the investigator. | |
| Grade 4: | Hospitalization may be indicated. Subject is | |
| Life-threatening; pressor or | permanently discontinued from further trial | |
| ventilatory support indicated | treatment administration. | |

Appropriate resuscitation equipment should be available in the room and a physician readily available during the period of drug administration.

For Further information, please refer to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE) at <a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>

Infusion Reactions

## 3.13 Follow-up to Resolution

Subjects should be followed to resolution. The Adverse Experience eCRF should be updated with information regarding duration and clinical course of the event. Information obtained from the consulting specialist, including diagnosis, should be recorded in the appropriate AE fields. Free-text fields should be used to record narrative information:

- Clinical course of the event
- Course of treatment
- Evidence supporting recovery

## - Follow-up to the clinical course

Any treatments administered for the event should also be entered in the Concomitant Medication eCRF.

**5.**Events of Clinical Interest (ECI) – Reference Table

| 3.Events of Chinear Interest (ECI) | tererence rubic | |
|---|---|---|
| Pneumonitis (reported as ECI if $\geq$ Gr | rade 2) | |
| Acute interstitial pneumonitis | Interstitial lung disease | Pneumonitis |
| Colitis (reported as ECI if ≥ Grade 2 | or any grade resulting in dose modific | cation or use of systemic steroids to treat |
| Intestinal Obstruction | Colitis | Colitis microscopic |
| Enterocolitis | Enterocolitis hemorrhagic | Gastrointestinal perforation |
| Necrotizing colitis | Diarrhea | |
| Endocrine (reported as ECI if ≥ Grade to treat—the AE) | e 3 or ≥ Grade 2 and resulting in dose i | nodification or use of systemic steroids |
| Adrenal Insufficiency | Hyperthyroidism | Hypophysitis |
| Hypopituitarism | Hypothyroidism | Thyroid disorder |
| Thyroiditis | Hyperglycemia, if ≥Grade 3 and asso | ociated with ketosis or metabolic acidosis |
| Endocrine (reported as ECI) | | |
| Type 1 diabetes mellitus (if new onset) | | |
| Hematologic (reported as ECI if $\geq$ Gr treat the AE) | rade 3 or any grade resulting in dose n | nodification or use of systemic steroids to |
| Autoimmune hemolytic anemia | Aplastic anemia | Thrombotic Thrombocytopenic Purpura (TTP) |
| Idiopathic (or immune) Thrombocytonenia Purpura (ITP) Any Grade 4 anemia regardless of under | Disseminated Intravascular Coagulation (DIC) lying mechanism | Haemolytic Uraemic Syndrome (HUS) |
| | | ation or use of systemic steroids to treat the |
| Hepatitis | Autoimmune hepatitis | Transaminase elevations (ALT and/or |
| Infusion Reactions (reported as ECI for | or any grade) | |
| Allergic reaction | Anaphylaxis | Cytokine release syndrome |
| Serum sickness | Infusion reactions | Infusion-like reactions |
| Neurologic (reported as ECI for any g | rade) | |
| Autoimmune neuropathy | Guillain-Barre syndrome | Demyelinating polyneuropathy |
| Myasthenic syndrome | | |
| Ocular (report as ECI if ≥ Grade 2 or | any grade resulting in dose modificati | ion or use of systemic steroids to treat the |
| Uveitis | Iritis | |
| Renal (reported as ECI if $\geq$ Grade 2) | • | |
| Nephritis | Nephritis autoimmune | Renal Failure |
| Renal failure acute | Creatinine elevations (report as ECI i modification or use of systemic steroid | f ≥Grade 3 or any grade resulting in dose ds to treat the AE) |
| Skin (reported as ECI for any grade) | , | |
| Dermatitis exfoliative | Erythema multiforme | Stevens-Johnson syndrome |
| Toxic epidermal necrolysis | | |
| Skin (reported as ECI if ≥ Grade 3) | • | |
| Skin (reputied as ECI II \(\text{Grade 3}\) | | |

| Pruritus | Rash | Rash generalized |
|---|---|---|
| Rash maculo-papular | | |
| Any rash considered clinically significant | nt in the physician's judgment | |
| Other (reported as ECI for any grade) | | |
| Myocarditis | Pancreatitis | Pericarditis |
| Any other Grade 3 event which is considered immune-related by the physician | | |

## 6. Past Medical History Related to Dermatologic Event

## **Past Medical History:**

Any preexisting conditions not previously reported (e.g., drug allergy) should be entered into the Medical History eCRF.

| 1. Do | bes the subject have any allergies? |
|---|---|
| | □ Yes □ No |
| If yes, | please obtain the following information: |
| | a. Any allergy to drugs (including topical or ophthalmic drugs)? |
| | □ Yes □ No |
| | List the drug name(s) and describe the type of allergic response (e.g. rash, anaphylaxis etc): |
| | b. Any allergy to external agents, such as laundry detergents, soaps, poison ivy, nickel, etc.? |
| | □Yes □ No |
| | Describe the agent and type of allergic response: |
| | c. Any allergy to food? □ Yes □ No |
| | Describe the food and type of allergic response: |
| | Any allergy to animals, insects? □ Yes □ No |
| | Describe the allergen and type of allergic response: |
| | Any other allergy? □ Yes □ No |
| | Describe the allergen and type of allergic response: |
| 2. Do | bes the subject have any other history of skin reactions, skin eruptions, or rashes? |

| If so what kind? |
|---|
| 3. Has the subject ever been treated for a skin condition? □ Yes □ No If so what kind? |
| 4. Is the current finding similar to a past experience? □ Yes □ No |
| 7. Presentation of the Dermatologic Event |
| Presentation of the event: |
| Collect information on clinical presentation and potential contributing factors. Key information should be summarized and entered on the Adverse Experience eCRF. Any treatments administered should be entered on the Concomitant Medication eCRF. |
| 1. What is the onset time of the skin reaction, skin eruption, or rash relative to dose of study drug? |
| 2. Has the subject contacted any known allergens? □ Yes □ No |
| If so what kind? |
| 3. Has the subject contacted new, special, or unusual substances (e.g., new laundry detergents, soap, personal care product, poison ivy, etc.)? $\square$ Yes $\square$ No |
| If so what kind? |
| <ul><li>4. Has the subject taken any other medication (over the counter, prescription, vitamins, and supplement)?</li><li>□ Yes □ No</li></ul> |
| If so what kind? |
| 5. Has the subject consumed unaccustomed, special or unusual foods? □ Yes □ No |
| If so what kind? |
| 6. Does the subject have or had in the last few days any illness? □ Yes □ No |
| If so what kind? |
| 7. Has the subject come into contact with any family or house members who are ill? $\Box$ Yes $\Box$ No |
| If so what kind? |
| 8. Has the subject recently been near children who have a skin reaction, skin eruption, or rash (e.g. Molluscum Contagiosum)? $\square$ Yes $\square$ No |
| 9. Has the subject had recent sun exposure? □ Yes □ No |
| 10. For the current rash, have there been any systemic clinical signs? □ Yes □ No |

| i. Anaphylaxis? □ Yes □ No | |
|---|---|
| ii. Signs of hypotension? □ Yes □ No | |
| iii. Signs of dyspnea? □ Yes □ No | |
| iv. Fever, night sweats, chills? □ Yes □ No | |
| 11. For the current rash, has the subject needed subcutaneous epinephrine or other system catecholamine therapy? $\square$ Yes $\square$ No | c |
| If so what kind? | |
| 12. For the current rash, has the subject used any other medication, such as inhaled bronchodilators, antihistaminic medication, topical corticosteroid, and/or systemic corticosteroid? □ Yes □ No | |
| List medication(s) and dose(s) | |
| 13. Is the rash pruritic (itchy)? □ Yes □ No | |
| 8. Focused Skin Examination | |
| Focused Skin Examination: | |
| Key information should be summarized and entered on the Adverse Experience eCRF. | |
| Key information should be summarized and entered on the Adverse Experience eCRF. Primary Skin Lesions Description | |
| Primary Skin Lesions Description | |
| Primary Skin Lesions Description Color: | |
| Primary Skin Lesions Description Color: | |
| Primary Skin Lesions Description Color: General description: | |
| Primary Skin Lesions Description Color: General description: | |
| Primary Skin Lesions Description Color: General description: Describe the distribution of skin reaction, skin eruption, or rash on the body: | |
| Primary Skin Lesions Description Color: General description: Describe the distribution of skin reaction, skin eruption, or rash on the body: | |